### **CLINICAL STUDY PROTOCOL**

**Protocol Number:** CA-ALT-803-02-13

A Study of ALT-803 in Patients with Relapsed or Refractory Multiple Myeloma **Protocol Title:** 

**Date of Protocol:** 

January 7, 2014 Version# 01

**Sponsor Contact:** Altor BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

## **Table of Contents**

| <b>3</b> | YNOPSI | IS | 6 |
|---|---|---|---|
| 1. | OBJ | ECTIVES | 12 |
| | 1.1 | Primary objectives | .12 |
| | 1.2 | SECONDARY OBJECTIVES | |
| 2. | | CKGROUND | |
| ۷. | 2.1 | ALT-803 – GENERAL INFORMATION | |
| | 2.1 | MULTIPLE MYELOMA | |
| | 2.2 | IMMUNE-BASED THERAPIES FOR CANCER | |
| | 2.3 | PHARMACOLOGICAL EFFECTS OF ALT-803 IN VITRO AND IN ANIMALS | |
| | 2.4.1 | Development of ALT-803 (IL-15N72D:IL-15RaSu/IgG1 Fc complex) | |
| | 2.4.2 | | |
| | 2.4.3 | | |
| | 2.4.4 | | |
| | 2.4.5 | Anti-myeloma mechanism of action of ALT-803 | 17 |
| | 2.5 | Non-clinical toxicology | |
| | 2.5.1 | <b>→</b> | |
| | 2.5.2 | , | |
| | | PHARMACOKINETICS | |
| | 2.6.1 | I | |
| | 2.6.2<br>2.7 | Clinical pharmacokinetics | |
| | 2.8 | HUMAN EXPERIENCE | |
| 3. | | TONALE FOR THE CURRENT STUDY | |
| 4. | OVE | ERALL STUDY DESIGN | 22 |
| 5. | STU | DY POPULATION | 24 |
| | 5.1 | INCLUSION CRITERIA | 24 |
| | 5.2 | EXCLUSION CRITERIA | 25 |
| | 5.3 | INCLUSION OF WOMEN AND MINORITIES | 25 |
| 6. | STU | DY DESIGN | 26 |
| | 6.1 | STUDY FLOW DIAGRAM | |
| | 6.2 | SCREENING AND ENROLLMENT | |
| | 6.3 | STUDY TREATMENT | - |
| | 6.3.1 | | |
| | 6.3.2 | | |
| | | Study drug preparation | 27 |
| | 6.3.4 | , 0 | |
| | 6.3.5 | 1 17 0 | |
| | 6.4 | DURATION OF PATIENT PARTICIPATION | 29 |
| | <i>( =</i> | | |
| | 6.5 | DOSE ESCALATION PHASE | 29 |
| | 6.6 | EXPANSION PHASE | 29<br>30 |
| | 6.6<br>6.7 | EXPANSION PHASE | 29<br>30 |
| | 6.6<br>6.7<br><i>6.7.1</i> | EXPANSION PHASE | 29<br>30<br>31 |
| | 6.6<br>6.7<br>6.7.1<br>6.7.2 | EXPANSION PHASE STOPPING RULES During dose escalation phase of the study During expansion phase of the study | 29<br>30<br>31<br><i>31</i> |
| | 6.6<br>6.7<br>6.7.1<br>6.7.2<br>6.7.3 | EXPANSION PHASE STOPPING RULES | 29<br>30<br>31<br>31 |
| | 6.6<br>6.7<br>6.7.1<br>6.7.2 | EXPANSION PHASE STOPPING RULES During dose escalation phase of the study During expansion phase of the study At any time during the study PATIENT MONITORING, RESPONSE EVALUATION, DISEASE PROGRESSION & SURVIVAL FOLLOW-UP | 29<br>30<br>31<br>31<br>31 |
| | 6.6<br>6.7<br>6.7.1<br>6.7.2<br>6.7.3<br>6.8 | EXPANSION PHASE STOPPING RULES | 29<br>30<br>31<br>31<br>31<br>32 |

| 6.9 | DOSE LIMITING TOXICITY | 32 |
|---|---|---|
| 6.9 | 9.1 Definition of dose limiting toxicity | 32 |
| 6.9 | 9.2 Definition of maximum tolerated dose (MTD) | 33 |
| 6.9 | 9.3 Definition of minimal efficacious dose (MED) | |
| 6.10 | STUDY TREATMENT DISCONTINUATION | 33 |
| 6. | 10.1 Study treatment discontinuation events | 33 |
| 6. | 10.2 Replacement of participants | 33 |
| 6 | 10.3 Follow-ups after treatment discontinuation | |
| | 6.10.3.1. Discontinuation due to SAEs or on-going study drug related AEs | 34 |
| | 6.10.3.2. Discontinuation due to any other reasons | |
| 6.11 | STUDY TREATMENT INTERRUPTION | 34 |
| 6 | 11.1 Kidney dysfunction | 34 |
| 6 | 11.2 Hematological dysfunction | |
| 6 | 11.3 Hypotension | |
| 6 | 11.4 Allergic reactions and cytokine release syndrome/acute infusion reaction | |
| 6.12 | | |
| 6. | 12.1 Hypotension and capillary leak syndrome | |
| | 12.2 Pulmonary dysfunction | |
| | 12.3 Impaired kidney and liver functions | |
| 6. | 12.4 Infection | |
| | 12.5 Fever and chills | |
| | 12.6 Gastritis | |
| 6. | 12.7 Diarrhea, nausea and vomiting | |
| 6. | 12.8 Pruritus and dermatitis | |
| | 12.9 Acidosis | |
| 6 | 12.10 Life-threatening toxicities | |
| 6 | 12.11 Other supportive care | |
| 6 | | |
| 0.1 | 12.12 Drug interaction | |
| 7. ST | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | 38 |
| 7. Si | FUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | <b>38</b> |
| 7. ST 7.1 7.2 | FUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 38<br>38 |
| 7. ST 7.1 7.2 7.3 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 38<br>38<br>38 |
| 7.1<br>7.2<br>7.3<br>7.4 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 38<br>38<br>38<br>38 |
| 7.1<br>7.2<br>7.3<br>7.4 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 38<br>38<br>38<br>38 |
| 7. ST 7.1 7.2 7.3 7.4 8. ST | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 38<br>38<br>38<br>38<br>39 |
| 7. \$7.1<br>7.2<br>7.3<br>7.4<br><b>8.</b> \$7.8 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 383838383839 |
| 7.1<br>7.2<br>7.3<br>7.4<br>8. \$1<br>8.1<br>8.2 | AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 38383838383939 |
| 7.1<br>7.2<br>7.3<br>7.4<br>8. ST<br>8.1<br>8.2<br>8.2 | AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 38383838393940 |
| 7.1 7.2 7.3 7.4 8. ST 8.1 8.2 8.2 8.2 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 38383839394040 |
| 7.1 7.2 7.3 7.4 8. ST 8.1 8.2 8.2 8.2 8.2 8.2 | AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 3838383939404040 |
| 7.1 7.2 7.3 7.4 8. ST 8.1 8.2 8.2 8.2 8.2 8.2 8.2 | AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 383838393940404040 |
| 7.1 7.2 7.3 7.4 8. \$1 8.2 8.2 8.2 8.2 8.2 8.2 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 38383839394040404040 |
| 7.1 7.2 7.3 7.4 8. ST 8.1 8.2 | AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY ACCOUNTABILITY PACKAGING LABELING | 3838383939404040404040 |
| 7.1 7.2 7.3 7.4 8. ST 8.1 8.2 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | 3838383939404040404040 |
| 7. ST<br>7.1<br>7.2<br>7.3<br>7.4<br>8. ST<br>8.1<br>8.2 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | 3838383939404040404040404040 |
| 7. \$7.1 7.2 7.3 7.4 8. \$7.8 8.1 8.2 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | 38383839404040404040404040404040404041 |
| 7. \$7.1 7.2 7.3 7.4 8. \$7.8 8.1 8.2 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | 3838383940404040404040404040404141 |
| 7.1 7.2 7.3 7.4 8. ST 8.1 8.2 | TUDY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | 38383839404040404040404040414141 |
| 7.1 7.2 7.3 7.4 8. ST 8.1 8.2 | AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY ACCOUNTABILITY PACKAGING LABELING FUDY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR. PROCEDURE AND TESTS 2.1 Assays for immune cell levels and phenotype 2.2 Medical history & prior therapy 2.3 Pregnancy test. 2.4 Physical examination 2.5 Vital signs, body weight & height 2.6 Cardiac assessment 2.7 Pulmonary function monitoring 2.8 Clinical blood tests 2.9 Disease assessment tests and procedures 2.10 Adverse event assessment 2.11 Response assessment 2.11 Response assessment 2.12 Disease progression and survival follow-up | 38383939404040404040414141 |
| 7. \$7.1 7.2 7.3 7.4 8. \$7.8 8.1 8.2 | AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING AVAILABILITY | 383839394040404040404141414142 |
| 7. \$7.1 7.2 7.3 7.4 8. \$7.8 8.1 8.2 | AVAILABILITY | 38383839404040404040414141414242 |
| 7. ST<br>7.1<br>7.2<br>7.3<br>7.4<br>8. ST<br>8.1<br>8.2 | AVAILABILITY | 38383839404040404040414141414242 |
| 7. ST<br>7.1<br>7.2<br>7.3<br>7.4<br>8. ST<br>8.1<br>8.2 | AVAILABILITY | 383839394040404040404141414141424243 |

| 9.2 | EFFECT ASSESSMENT SCHEDULE | 43 |
|---|---|---|
| 9.3 | METHODOLOGY OF RESPONSE EVALUATION | |
| 9.4 | RESPONSE EVALUATION CRITERIA | 42 |
| 9.5 | DISEASE PROGRESSION EVALUATION CRITERIA | 45 |
| 10. | STATISTICAL ANALYSIS | 46 |
| 10.1 | STUDY OBJECTIVES | |
| 10.2 | SAMPLE SIZE | |
| 10.3 | DATA COLLECTION | |
| 10.4 | Data analysis | |
| 10. | 4.1 Analysis of safety | |
| - 0 - | 4.2 Analysis of response | 47 |
| 10. | 4.3 Pharmacokinetics | 47 |
| <b>11.</b> 1 | REGULATORY AND REPORTING REQUIREMENTS | 48 |
| 11.1 | ADVERSE EVENTS RECORDING, REPORTING AND COMMUNICATION | 48 |
| 11.2 | ADVERSE EVENT TERMINOLOGY AND DEFINITIONS | 48 |
| 11.3 | ADVERSE EVENT REPORTING PROCEDURES | 49 |
| 11.4 | ADVERSE EVENT EXPEDITED REPORTING GUIDELINES | 50 |
| 11.5 | SUBMISSION OF SERIOUS ADVERSE EVENT REPORTING | 50 |
| 11.6 | DATA REPORTING FORMS | 50 |
| 11.7 | REPORT /DATA SUBMISSION ADDRESS & CONTACT | |
| 11.8 | PATIENT RECORDS, QUALITY ASSURANCE, RECORDS RETENTION | 51 |
| 11.9 | METHOD OF REVIEW | 51 |
| 11.10 | SPECIAL REGULATORY CONSIDERATIONS | 52 |
| | 10.1 HIPAA | |
| | 10.2 Protocol amendments, informed consent, and IRB approval | |
| 12. | CONFIDENTIALITY | 52 |
| 13. | ETHICAL STANDARDS & INVESTIGATOR OBLIGATIONS | 52 |
| 14. | LIST OF EXPECTED ADVERSE EVENTS | 53 |
| 15. | CTCAE | 55 |
| REFER | ENCES | 50 |
| APPEN | DIX A: ECOG | 58 |
| APPEN | DIX B: NEW YORK HEART ASSOCIATION CLASSIFICATION | 5 |
| | DIX C: ETHICAL STANDARDS | |
| | DIX D: INVESTIGATOR OBLIGATIONS | |
| | DIX E: CONTACT LIST - ALTOR | |
| | DIX F: CONTACT LIST - DATA SAFETY MONITORING BOARD (DSMB) | |
| | DIX G: CONTACT LIST - DATA SAFETT MONTORING BOARD (DSMB) | |
| | V1/1 V: VV: 1.1/1 V I LID I = L//IDVIV/1 VINI/D::::::::::::::::::::::::::::::::::: | |

#### **SYNOPSIS**

**Sponsor:** Altor Bioscience Corporation

**Protocol#:** CA-ALT-803-02-13

Study Drug Name: Not applicable

**Study Treatment** 

Active agents: ALT-803, a "recombinant human super agonist interleukin-15 (IL-15) complex"

(AKA, IL-15N72D:IL-15RαSu/IgG1 Fc complex)

**Study Type:** Interventional

Study Phase: Ib/II

**Protocol Title:** A Study of ALT-803 in Patients with Relapsed or Refractory Multiple Myeloma

**Objectives:** To evaluate the safety and tolerability of escalating doses, identify the Maximum

Tolerated Dose level (MTD) or Minimum Efficacious Dose (MED) and designate a dose level for Phase II study (RP2D) of ALT-803 in patients with relapsed or

refractory multiple myeloma.

To evaluate the effect of ALT-803 on the peripheral absolute lymphocyte counts (ALC) and white blood cell (WBC) counts, the number and phenotype of

peripheral blood T (total and subsets) and NK cells.

To estimate the anti-tumor activity of ALT-803 by radiologic or pathologic disease

response, progression free survival, and overall survival in treated patients.

To characterize the immunogenicity and pharmacokinetic profile, including serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ and TNF-α, of ALT-803 in treated

patients.

**Study Design:** 

This is a Phase Ib/II, open-label, multi-center, competitive enrollment and dose-escalation study of ALT-803 in patients with relapsed or refractory multiple

myeloma.

The study includes a dose escalation phase to determine the MTD or MED using a modified classic (3+3) dose escalation design and to designate a dose level for the Phase II expansion phase (RP2D) and a two-stage expansion phase at the RP2D using a Simon two-stage design. In Phase I, five dose levels will be evaluated. A step-down dose level (cohort# -1) will be provided in the event of encountering DLT in two patients at the planned initial dose level. In the absence of unacceptable toxicity or disease progression, each enrolled patient will receive up to four 6-week study treatment cycles, each consisting of a 4-week treatment period and a 2-week rest period. In each cycle, patients will receive four doses of ALT-803 by intravenous injection weekly for 4 weeks followed by a 2-week rest period. Patients with sufficient recovery of toxicities from the previous treatment cycles will be eligible to continue study treatment. After receiving two treatment cycles, patients who have at least stable disease assessed at week 11-12 may receive up to two additional study treatment cycles followed by reassessment for continued tumor response.

January 7, 2014

The study will be conducted in conformity with Good Clinical Practice (GCP).

### **Treatments:**

The study treatment plan for each enrolled patient includes up to four 6-week study treatment cycles. In each cycle, patients will receive four weekly doses of ALT-803 by intravenous injection followed by a 20-day rest period. The rest period may be extended to include up to four additional weeks if necessary. Patients who do not experience or who sufficiently recover from toxicities of the previous treatment cycles will be eligible to continue the treatment included in the study treatment plan.

Treated patients will have up to two anti-tumor evaluation visits. Patients who receive at least three study drug doses during the first 2-cycle treatment period will be evaluated for anti-tumor response during week 11-12. Patients who have at least stable disease from the first anti-tumor evaluation and who meet other criteria to continue study treatment will receive up to two additional study treatment cycles, with the same treatment schedule and at the same dose level as the first two cycles, followed by reassessment for continued tumor response.

The study treatment and response evaluation schedule is illustrated below:

| Treatment Cycle | | Сус | le #1 | | REST | Cycle #2 | | | | Response<br>Evaluation | 1 ( VCIE #3 | | | | | Cycle #4 | | | | Response<br>Evaluation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Week | reatment Week 1 2 3 4 5-6 | | | | 7 | 8 | 9 | 10 | 11-12 | 13 | 14 | 15 | 16 | 17-18 | 19 | 20 | 21 | 22 | 23-24 | |
| Treatment Day | tment Day 1 8 15 22 23- | | 23-42 | 43 50 57 64 | | | 64 | 65-84 | 85 | 92 99 | | 106 | 107-126 | 127 | 134 | 141 | 148 | 149-168 | | |
| Dose# | 1 | 2 | 3 | 4 | | 5 | 6 | 7 | 8 | | 9 | 10 | 11 | 12 | | 13 | 14 | 15 | 16 | |
| Response Evaluation | | | | | Rest<br>weeks | | | | | X | | | | | Rest<br>weeks | | | | | X |
| ALT-803 | | X | X | X | | X | X | X | X | | X | X | X | X | | X | X | X | X | |

There are no restrictions on further therapies, such as chemotherapy, radiation therapy or surgery to be used after the protocol-specified therapy. Clearly, poststudy treatments could be of significant clinical benefit in selected patients, and these patients will be followed for outcome.

Enrolled patients will receive the study treatment at qualified cancer treatment centers with adequate diagnostic and treatment facilities to provide appropriate management of therapy and complications. ALT-803 will be administered by intravenous infusion into a central or peripheral vein under the supervision of a qualified physician experienced in the use of biologic anti-cancer agents.

### **Dose Escalation** Phase:

A modified 3 + 3 design will be used for identifying a tolerable dose for phase II studies by monitoring patients for DLTs to determine the MTD and for identifying an efficacious dose by monitoring patients' ALC and WBC count to determine the MED during the DLT observation period. The dose escalation phase is concluded when either the MTD or the MED is determined. A dose level (RP2D) will then be designated for Phase II study. There are five escalating dose levels of ALT-803 and a step-down cohort (-1) with a lower dose level of ALT-803 in the event that unexpected toxicity is encountered at the initial dose level.

Below are the planned dose levels of the study drug during the dose escalation phase of the study.

| Cohort | ALT-803 Dose (µg/kg) | Number of patients |
|-------------|----------------------|--------------------|
| -1 | 0.5 | 3 to 6 |
| 1 (initial) | 1 | 3 to 6 |
| 2 | 3 | 3 to 6 |
| 3 | 6 | 3 to 6 |
| 4 | 10 | 3 to 6 |
| 5 | 20 | 3 to 6 |

Dose limiting toxicity (DLT) is defined as follows: any study drug related toxicity that is of Grade 3 and does not resolve to Grade 1 or lower within a week despite the use of medical intervention or that is of Grade 4, with exceptions described in the study protocol.

The DLT Observation Period is defined as the duration of the first treatment cycle.

Maximum Tolerated Dose level (MTD) is defined as a dose level at which <2 out of 6 patients experienced DLT and that is one level below a dose that was not tolerated.

Minimal Efficacious Dose (MED) is defined as a dose level which produces an ALC  $\geq$ 25,000/µL sustained for 14 days or a total WBC  $\geq$ 35,000/µL sustained for 14 days among 2/3 or 4/6 of patients. For safety, we have also defined an "exceeding MED" as the occurrence of ALC  $\geq$ 35,000/µL or WBC  $\geq$ 50,000/µL sustained for 14 days.

# **Expansion Phase**

The two-stage expansion phase at the MTD or the MED level will be conducted using an optimal Simon's two-stage design. Objective response (OR) (defined as complete response (CR) + partial response (PR)) will be evaluated and set thresholds of lack of efficacy (OR rate (ORR) = 10%) and an efficacy level of interest (ORR = 30%) will be selected.

### **Stopping Rules:**

Patient enrollment will be temporarily suspended based on occurrence of any of the following events, and the study committee, including the sponsor, the Data Safety Monitoring Board and principal investigators will meet to discuss how to proceed with future patient enrollment in the study.

During the dose escalation phase of the study,

 If the maximum planned dose level has been reached, but neither the MTD nor MED can be determined. • If de-escalation occurs and the step-down dose level cannot be designated as the MTD or MED.

Any time during the expansion phase of the study,

CONFIDENTIAL

- More than 33% of patients experience a possible, probable or definite study drug related DLT.
- Favorable anti-tumor response data collected from enrolled patients.

At any time during the study,

The study committee may meet to discuss how to proceed with the study and may make any or all of the following recommendations for further patient enrollment:

- Downward adjust the study drug dose.
- Adjust the study drug dosing schedule.
- Recommend more effective pre-therapy, intra-therapy and post-therapy side effect mitigation interventions.
- Correct protocol technical errors that caused unnecessary dose omissions or premature treatment discontinuations. After correction of protocol errors, the DSMB may meet to re-evaluate the safety profile of the study treatment and recommend how to proceed with the study, if necessary.

### **Evaluations:**

Patients will be evaluated for clinical toxicities during the treatment. Patients' blood samples will be collected to assess the pharmacokinetic profile and immunogenicity of the study drug. The anti-tumor response will be evaluated at week 11-12 and week 23-24 from the start of study treatment. All patients who receive at least 3 doses of the study drug ALT-803 will be included in the anti-tumor response evaluation.

### Population:

Patients of 18 years of age and above with relapsed or refractory multiple myeloma. Patients also need to have adequate cardiac, pulmonary, liver and kidney functions and have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

### **Sample Size:**

A total of up to 30 assessable patients will be accrued to the dose escalation phase of the study (Phase Ib). Anticipated enrollment to this phase is 18 patients. Up to an additional 23 assessable patients will be enrolled at the expansion phase (Stage 1 and 2) of the study (Phase II). A total of approximately 41 assessable patients will be enrolled to complete the study. Assuming a 20% rate of ineligible or non-assessable cases, a total of up to 50 patients may be accrued to the study.

# Primary Endpoints

For Phase Ib only

(1) Determination of the MTD or MED and designation of the recommended dose level (RP2D) for Phase II study of ALT-803 in patients with relapsed or refractory multiple myeloma.

### For Phase Ib & II

- (2) Safety profile of ALT-803 in treated patients.
- (3) Disease response rate of treated patients.

### **Secondary**

### **Endpoints**

- (1) Evaluation of the effect of ALT-803 on the peripheral ALC and WBC counts, the number and phenotype of peripheral blood T (total and subsets) and NK cells in treated patients.
- (2) Duration of response in treated patients.
- (3) Progression free survival of treated patients.
- (4) Overall survival of treated patients.
- (5) Characterization of the immunogenicity and pharmacokinetic profile, including serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ and TNF-α, of ALT-803 in treated patients.

## Pharmacokinetics & Biomarkers:

Fresh blood samples will be collected to assess immune cell levels and phenotype, and serum samples for pharmacokinetics, immunogenicity of the study drug ALT-803, and the serum levels of IL-2, IL-4, IL-6, IL-10, IFN- $\gamma$  and TNF- $\alpha$  after ALT-803 administration in treated patients. Blood samples for pharmacokinetic analysis will be taken on the first day of ALT-803 administration in the first study treatment cycle. Venous blood will be obtained at Time 0 (before the start of infusion), at 30 minutes, and 2, 4, 6 and 24 hours from Time 0 for the assessment of ALT-803 serum concentrations. Non-compartmental and compartmental analyses will be conducted. In addition, the same blood samples collected for PK analysis will be used to assess the serum levels of IL-2, IL-4, IL-6, IL-10, IFN- $\gamma$  and TNF- $\alpha$ . Fresh blood samples for immune cell levels and phenotype testing will be collected before the start of first and fourth dose of study drug infusion in each treatment cycle. Bone marrow samples will be collected for future analysis of molecular markers associated with responses or resistance to ALT-803 in patients with relapsed or refractory multiple myeloma.

### **Monitoring Tests:**

Blood samples for standard chemistry and CBC with differential will be obtained at screening, on each study drug infusion day, and at follow-up visits. Blood samples for immunogenicity testing for anti-ALT-803 antibodies will be collected prior to dosing on the first ALT-803 infusion day and at weeks 7 and 12 from the initial dose of study treatment. Blood and urine samples will be collected on each follow-up visit for response assessment.

## Response Assessment:

There are at least two response assessments for treated patients: the first assessment during week 11-12 and the second assessment during week 23-24 from the start of study treatment. After completion of the first two cycles of study treatment, patients who have received at least 3 doses of study drug will have the first response assessment. After completion of the two additional cycles of study treatment, patients, regardless of the number of additional study drug doses received, will have the second response assessment. Response assessments will be carried out according to the new International Uniform Response Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. Baseline evaluations should be performed up to 14 days before study treatment starts.

# Progression & Survival

CA-ALT-803-02-13 Version# 01 January 7, 2014

**Assessment:** 

Progression-free survival, overall survival, and duration of response of all treated patients will be assessed every three months during year 1 and then every 6 months during years 2 and 3 from the start of study treatment, or through the point designated as the end of the study follow up.

**Adverse Events:** 

All patients will be monitored and evaluated for clinical toxicities during the treatment period and queried at each follow-up visit for Adverse Events (AEs). Patients may volunteer information concerning AEs. All adverse events will be graded by using the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0), and logged in the patient Case Report Form. The study centers should report all Serious Adverse Events (SAEs) and all events that trigger patient's study treatment discontinuation to the sponsor via phone, fax or email (or a combination) no more than 24 hours after learning of the event. The sponsor will use the information to manage and coordinate the dose escalation, cohort expansion and patient enrollment. The sponsor will then inform all of the participating clinical sites of the current dose level and the number of patients to be enrolled at that level, or of any patient enrollment suspension via phone, fax or email within 24 hours of learning of the event. The study centers should report all other adverse events to the sponsor following the guidelines defined in the study protocol. All study drug related AEs that are both serious and unexpected will be reported to the FDA in an expedited manner in accordance with 21 CFR §312.32.

**Statistical Plan:** 

For each cohort, all AEs will be tabulated and examined and all safety, pharmacokinetic and tumor response data will be evaluated. For estimation of duration of response and progression free survival, the Kaplan-Meier method will be used. P-values of  $\leq 0.05$  (two-sided) will be considered to indicate statistical significance.

### 8. STUDY CALENDAR, CLINICAL PROCEDURES & TESTS

### 8.1 Study calendar

| TESTS & PROCEDURES | SCREEN/<br>BASELINE <sup>1</sup> | Т | REAT | | | REST | | REAT:<br>CYCL | | Γ | 1 <sup>ST</sup> RESPONSE<br>ASSESSMENT | TREATMENT CYCLES<br>#3 AND #4 | 2 <sup>ND</sup> RESPONSE<br>ASSESSMENT | FOLLOW-UPS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | | | | 1 | | | | 7 8 9 10 | | 3 | 4-5 | 6 | 9 12 18 24 30 36 | |
| Study Week | | 1 | 2 | 3 | 4 | 5-6 | 7 | | | 11-12 | 13-22 | 23-24 | | |
| Study Day | | 1 | 8 | 15 | 22 | 23-42 | 43 | 50 | 57 | 64 | 65-84 | 85-148 | 149-168 | Any day during the month |
| Tolerance Window | | | +/- 2 | days | | 23-42 | | +/- 2 | lays | | Any day | | Any day | |
| Medical history | X | | | | | | | | | | | | | |
| Serum pregnancy test <sup>2</sup> | X | | | | | | | | | | | Follow Institution's | | |
| Complete physical exam | X | X | | | | | X | | | | X | standard of care (SOC) | X | |
| Vital signs, Weight, Height <sup>3</sup> , Cardiac & Lung function monitoring | X | X | X | X | X | | X | X | X | X | X | policy. If performed, follow the | X | |
| Concurrent medication | X | X | X | X | X | | X | X | X | X | X | same schedule as in the | X | |
| Adverse event assessment <sup>4</sup> | X | X | X | X | X | | X | X | X | X | X | first two cycles of study | X | |
| CBC with Differential | X | X | X | X | X | R | X | X | X | X | X | treatment. | X | |
| Blood Chemistry | X | X | X | X | X | E | X | X | X | X | X | | X | |
| EKG | X | $X^5$ | | | | | X | | | | | | | |
| PFT only when clinically indicated | X | | | | | S | | | | | | | | |
| Response evaluation <sup>6</sup> | | | | | | T | | | | | X | | X | |
| Serum quantitative immunoglobulins | X | | | | | | | | | | X | | X | |
| SPEP | X | | | | | P | | | | | X | | X | |
| UPEP-random | X | | | | | _ | | | | | X | | X | |
| SIFE | X | | | | | E | | | | | X | | X | |
| UIFE -random | X | | | | | R | | | | | X | | X | |
| Serum FLC assay <sup>6.1</sup> | X | | | | | | | | | | X | | X | |
| Bone marrow plasma cell percentage <sup>6.2</sup> | X | | | | | I | | | | | X | | X | |
| Bone marrow immunohistochemistry or immunofluorescence <sup>6.3</sup> | | | | | | 0 | | | | | X | | X | |
| Soft tissue plasmacytomas assessment <sup>6,4</sup> | | | | | | R | | | | | X | | X | |
| Disease & survival follow-up/post-therapies <sup>7</sup> | | | | | | - 1 | | | | | | | | x x x x x x |
| Immune cell levels & phenotype <sup>8,11</sup> | | $X^8$ | | | $X^8$ | | $X^8$ | | | $X^8$ | | | | |
| PK <sup>x</sup> , IL-2, IL-4, IL-6, IL-10, IFN-γ, TNF-α <sup>9,11</sup> | | X <sup>9</sup> | | | | | | | | | | | | |
| Immunogenicity tests <sup>10, 11</sup> | | $X^{10}$ | | | | | X | | | | X | | | |
| Study drug (ALT-803) | | a1 | a2 | а3 | a4 | | a5 | a6 | a7 | a8 | | Follow the same schedule as in the first 2 cycles of study treatment | | |

Screening/baseline evaluations are performed ≤ 14 days prior to start of therapy. If the patient's condition is deteriorating, ECOG status and laboratory evaluations should be repeated within 48 hours initiation of study treatment infusion. Pregnancy test is for women with childbearing potential only. Vital signs (especially blood pressure), clinical status and laboratory tests should be reviewed before start of therapy. Vital signs will be evaluated at 15, 30, 60 and 120 minutes and then hourly post infusion until discharge (or at completion of dose monitoring) from the clinic, and body weight before infusion on drug infusion day. Patients who have an on-going study drug-related SAE upon study completion or at discontinuation of study will be contacted by the investigator or his/her designee every week until the event is resolved or determined to be irreversible. If the screening EKG was performed within 14 days prior to start of study treatment, the EKG is not required. Disease response and progression assessment will be evaluated using the new International Uniform Response Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. Uniform Response Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. Uniform Protein are unmeasurable. Only when serum and urine M-protein are unmeasurable and bone marrow plasma cell percentage > 30% at baseline. Only when scR is to be determined. Uniform Response Criteria for Protein are unmeasurable and bone marrow plasma cell percentage > 30% at baseline. Uniform Response Criteria for Multiple Myeloma Working Group. Uniform Response Criteria for Multiple Myeloma Visual Myeloma Working Group. Uniform Response Criteria

### **CLINICAL STUDY PROTOCOL**

CA-ALT-803-02-13 **Protocol Number:** 

A Study of ALT-803 in Patients with Relapsed or Refractory Multiple Myeloma **Protocol Title:** 

**Date of Protocol:** 

January 7, 2014 Version# 01 Version# 02 February 3, 2014

**Sponsor Contact:** Altor BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

## **Table of Contents**

| 5 | NOPSI | | 6 |
|---|---|---|---|
| 1. | OBJ | ECTIVES | 12 |
| | 1.1 | PRIMARY OBJECTIVES | . 12 |
| | 1.2 | SECONDARY OBJECTIVES | – – |
| 2. | RAC | KGROUND | |
| | 2.1 | ALT-803 – General information | |
| | 2.1 | MULTIPLE MYELOMA | |
| | 2.3 | IMMUNE-BASED THERAPIES FOR CANCER | |
| | 2.4 | PHARMACOLOGICAL EFFECTS OF ALT-803 IN VITRO AND IN ANIMALS | |
| | 2.4.1 | Development of ALT-803 (IL-15N72D:IL-15RaSu/IgG1 Fc complex) | |
| | 2.4.1 | In vitro biological activity of ALT-803 | |
| | 2.4.3 | In vivo biological activity of ALT-803 | |
| | 2.4.4 | Potent anti-tumor activity of ALT-803 in mouse models | |
| | 2.4.5 | Anti-myeloma mechanism of action of ALT-803 | |
| | 2.5 | Non-clinical toxicology | |
| | 2.5.1 | Multi-dose toxicity studies in mice | 17 |
| | 2.5.2 | Multi-dose toxicity studies in cynomolgus monkeys | 18 |
| | 2.6 | PHARMACOKINETICS | |
| | 2.6.1 | | |
| | 2.6.2 | $\mathbf{I}$ | |
| | 2.7 | RATIONALE FOR HUMAN CLINICAL STARTING DOSE. | |
| | 2.8 | HUMAN EXPERIENCE | 20 |
| 3. | RAT | TONALE FOR THE CURRENT STUDY | 21 |
| 4. | OVE | RALL STUDY DESIGN | 22 |
| 5. | | DY POPULATION | |
| • | 5.1 | INCLUSION CRITERIA | |
| | 5.2 | EXCLUSION CRITERIA. | |
| | 5.3 | INCLUSION OF WOMEN AND MINORITIES. | |
| , | | | |
| 6. | | DY DESIGN | |
| | 6.1 | STUDY FLOW DIAGRAM | |
| | 6.2 | SCREENING AND ENROLLMENT | |
| | 6.3 | STUDY TREATMENT | |
| | 6.3.1 | | |
| | 6.3.2 | Treatment regimen and study scheme | |
| | 6.3.3 | Study drug preparation | |
| | 6.3.4<br>6.3.5 | Study drug administration | |
| | 6.4 | Pre and post-therapy intervention guidelines DURATION OF PATIENT PARTICIPATION | |
| | 6.5 | DOSE ESCALATION PHASE | |
| | 6.6 | EXPANSION PHASE | |
| | 6.7<br>6.7.1 | STOPPING RULES | |
| | 6.7.2 | During aose escalation phase of the study During expansion phase of the study | |
| | 6.7.3 | At any time during the study | |
| | 6.8 | PATIENT MONITORING, RESPONSE EVALUATION, DISEASE PROGRESSION & SURVIVAL FOLLOW-UP | |
| | 6.8.1 | Patient monitoring | |
| | 6.8.2 | Response evaluation. | |
| | 6.8.3 | Disease progression and survival follow-up | |

| | 6.9 I | OSE LIMITING TOXICITY | |
|---|---|---|---|
| | 6.9.1 | Definition of dose limiting toxicity | |
| | 6.9.2 | Definition of maximum tolerated dose (MTD) | |
| | 6.9.3 | Definition of minimal efficacious dose (MED) | |
| | 6.10 | TUDY TREATMENT DISCONTINUATION | |
| | 6.10.1 | Study treatment discontinuation events | |
| | 6.10.2 | Replacement of participants | |
| | 6.10.3 | Follow-ups after treatment discontinuation | |
| | | 0.3.1. Discontinuation due to SAEs or on-going study drug related AEs | |
| | | 0.3.2. Discontinuation due to any other reasons | |
| | 6.11 | TUDY TREATMENT INTERRUPTION | |
| | 6.11.1 | Kidney dysfunction | |
| | 6.11.2 | Hematological dysfunction | |
| | 6.11.3 | Hypotension | |
| | 6.11.4 | Allergic reactions and cytokine release syndrome/acute infusion reaction | |
| | | GENERAL SUPPORTIVE CARE GUIDELINES AND DRUG INTERACTION | |
| | 6.12.1 | Hypotension and capillary leak syndrome | |
| | 6.12.2 | Pulmonary dysfunction | |
| | 6.12.3 | Impaired kidney and liver functions | |
| | 6.12.4 | Infection | |
| | 6.12.5 | Fever and chills | |
| | 6.12.6 | Gastritis | |
| | 6.12.7 | Diarrhea, nausea and vomiting | |
| | 6.12.8 | Pruritus and dermatitis | |
| | 6.12.9 | Acidosis | |
| | 6.12.10<br>6.12.1 | , e | |
| | 6.12.12 | •• | |
| | 0.12.12 | Drug interaction | |
| 7 | CTHE | V DDIIC, AVAII ADII ITV ACCOUNTADII ITV DACKACING & LADEI INC | |
| 7. | | Y DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | 38 |
| 7. | 7.1 | AVAILABILITY | 38 |
| 7. | 7.1 A | AVAILABILITYACCOUNTABILITY | 38<br>38 |
| 7. | 7.1 A<br>7.2 A<br>7.3 I | AVAILABILITYACCOUNTABILITY | 38<br>38<br>38 |
| 7. | 7.1 A<br>7.2 A<br>7.3 I | AVAILABILITYACCOUNTABILITY | 38<br>38<br>38 |
| | 7.1 7.2 7.3 I 7.4 I | AVAILABILITY | 38<br>38<br>38 |
| 7.<br>3. | 7.1 A<br>7.2 A<br>7.3 I<br>7.4 I<br>STUD | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING PY CALENDAR, CLINICAL PROCEDURES & TESTS | |
| | 7.1 7.2 7.3 II 7.4 II STUD 8.1 55 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING ACKAENDAR, CLINICAL PROCEDURES & TESTS | |
| | 7.1 7.2 7.3 II 7.4 II STUD 8.1 5.8.2 II | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING LABELING STUDY CALENDAR, CLINICAL PROCEDURES & TESTS CRUCK TESTS PROCEDURE AND TESTS | |
| | 7.1 7.2 7.3 1.7.4 1.7.4 1.5 STUD 8.1 5.8.2 1.8.2.1 | AVAILABILITY ACCOUNTABILITY PACKAGING PACKAGING PABELING PASSED TESTS PROCEDURES & TESTS PROCEDURE AND TESTS Assays for immune cell levels and phenotype | 38<br>38<br>38<br>38<br>38<br>39<br>40 |
| | 7.1 7.2 7.3 17.4 17.4 17.4 17.4 18.1 18.2 18.2.1 8.2.2 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING ABELING TUDY CALENDAR, CLINICAL PROCEDURES & TESTS TUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy | 38<br>38<br>38<br>38<br>39<br>39<br>40<br>40 |
| | 7.1 7.2 7.3 17.4 17.4 17.5 STUE 8.1 8.2 18.2.2 8.2.3 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING ABELING BY CALENDAR, CLINICAL PROCEDURES & TESTS BY CALENDAR BY CALE | 38 38 38 39 40 40 40 40 |
| | 7.1 7.2 7.3 17.4 17.4 17.5 STUE 8.1 8.2.1 8.2.2 8.2.3 8.2.4 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING ABELING BY CALENDAR, CLINICAL PROCEDURES & TESTS CTUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination | 38 38 38 39 39 40 40 40 40 40 |
| | 7.1 7.2 7.3 1.7.4 1. STUE 8.1 5.2.1 8.2.2 8.2.3 8.2.4 8.2.5 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING ABELING BY CALENDAR, CLINICAL PROCEDURES & TESTS BTUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height | 38 38 38 39 40 40 40 40 40 40 |
| | 7.1 7.2 7.3 F. 7.4 F. STUD 8.1 8.2 F. 8.2.1 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING ABELING TUDY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment | 38 38 38 39 40 40 40 40 40 40 40 |
| | 7.1 7.2 7.3 F. 7.4 F. STUD 8.1 S.2 F. 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 | AVAILABILITY ACCOUNTABILITY ACKAGING ABELING ABELING TUDY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring | 38 38 38 39 40 |
| | 7.1 7.2 7.3 1.7.4 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING PY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring Clinical blood tests | 38 38 38 39 40 |
| | 7.1 7.2 7.3 F. 7.4 F. STUD 8.1 S.2 F. 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING BY CALENDAR, CLINICAL PROCEDURES & TESTS ASTUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring Clinical blood tests Disease assessment tests and procedures | 38 38 38 38 39 40 |
| | 7.1 7.2 7.3 7.4 7.4 7.4 7.4 7.4 7.5 8.1 8.2 8.2.1 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 8.2.8 8.2.9 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING PY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring Clinical blood tests | 38 38 38 38 39 40 |
| | 7.1 7.2 7.3 1.7.4 1.7.4 1.7.4 1.7.4 1.7.5 1.7.4 1.7.5 1.7.4 1.7.5 1.7.4 1.7.5 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING Y CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring Clinical blood tests Disease assessment tests and procedures Adverse event assessment | 38 38 38 38 38 39 40 |
| | 7.1 7.2 7.3 1.7.4 1.7.4 1.7.4 1.7.4 1.7.4 1.7.5 1.7.4 1.7.5 1.7.4 1.7.5 1.7.4 1.7.5 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING Y CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test. Physical examination Vital signs, body weight & height Cardiac assessment. Pulmonary function monitoring Clinical blood tests Disease assessment tests and procedures Adverse event assessment Response assessment | 38 38 38 39 40 |
| | 7.1 7.2 7.3 1.7.4 1.7.4 1.7.4 1.7.4 1.7.5 1.7.4 1.7.5 1.7.4 1.7.5 1.7.4 1.7.5 | AVAILABILITY | 38 38 38 38 39 40 40 40 40 40 41 |
| | 7.1 7.2 7.3 1.7.2 7.3 1.7.4 1.7.4 1.7.5 1.7.4 1.7.5 1.7.4 1.7.5 1. | AVAILABILITY ACCOUNTABILITY ACCAGING ABELING ABELING BY CALENDAR, CLINICAL PROCEDURES & TESTS BY CALENDAR BY CALENDAR BY COCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring Clinical blood tests Disease assessment tests and procedures Adverse event assessment Response assessment Disease progression and survival follow-up Pharmacokinetic (PK) testing | 38 38 38 38 39 40 40 40 40 40 41 |
| | 7.1 7.2 7.3 1.4 7.2 7.3 1.5 7.4 1.5 STUD 8.1 8.2.1 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 8.2.8 8.2.9 8.2.10 8.2.11 8.2.12 8.2.13 8.2.14 8.2.15 | AVAILABILITY ACCOUNTABILITY ACKAGING ABELING BELING ABELING ABELING ASELING ASELING BY CALENDAR, CLINICAL PROCEDURES & TESTS BY CALENDAR B | 38 38 38 38 38 39 40 |

| 9.2 EFFECT ASSESSMENT SCHEDULE | | 43 |
|---------------------------------------|-------------------------------|----|
| 9.3 METHODOLOGY OF RESPONSE EVALU | JATION | 43 |
| 9.4 RESPONSE EVALUATION CRITERIA | | 44 |
| 9.5 DISEASE PROGRESSION EVALUATION | CRITERIA | 45 |
| 10. STATISTICAL ANALYSIS | | 46 |
| 10.1 STUDY OBJECTIVES | | 46 |
| 10.2 SAMPLE SIZE | | 46 |
| 10.3 DATA COLLECTION | | 46 |
| 10.4 Data analysis | | 46 |
| 11. REGULATORY AND REPORTING | REQUIREMENTS | 48 |
| 11.1 ADVERSE EVENTS RECORDING, REPO | RTING AND COMMUNICATION | 48 |
| | DEFINITIONS | |
| 11.3 ADVERSE EVENT REPORTING PROCE | DURES | 49 |
| | TING GUIDELINES | |
| 11.5 SUBMISSION OF SERIOUS ADVERSE EV | VENT REPORTING | 50 |
| | S & CONTACT | |
| | NCE, RECORDS RETENTION | |
| | ATIONS | |
| · | onsent, and IRB approval | |
| | TIGATOR OBLIGATIONS | |
| 14. LIST OF EXPECTED ADVERSE EV | VENTS | 53 |
| 15. CTCAE | | 55 |
| REFERENCES | | 56 |
| APPENDIX A: ECOG | | 58 |
| APPENDIX B: NEW YORK HEART ASSO | CIATION CLASSIFICATION | 58 |
| | TIONS | |
| | AFETY MONITORING BOARD (DSMB) | |
| | ` ' | |
| APPENDIA G. CONTACT LIST - LABORA | ATORIES | 65 |

#### **SYNOPSIS**

**Sponsor:** Altor Bioscience Corporation

**Protocol#:** CA-ALT-803-02-13

Study Drug Name: Not applicable

**Study Treatment** 

Active agents: ALT-803, a "recombinant human super agonist interleukin-15 (IL-15) complex"

(AKA, IL-15N72D:IL-15RαSu/IgG1 Fc complex)

**Study Type:** Interventional

Study Phase: Ib/II

**Protocol Title:** A Study of ALT-803 in Patients with Relapsed or Refractory Multiple Myeloma

**Objectives:** To evaluate the safety and tolerability of escalating doses, identify the Maximum

Tolerated Dose level (MTD) or Minimum Efficacious Dose (MED) and designate a dose level for Phase II study (RP2D) of ALT-803 in patients with relapsed or

refractory multiple myeloma.

To evaluate the effect of ALT-803 on the peripheral absolute lymphocyte counts (ALC) and white blood cell (WBC) counts, the number and phenotype of

peripheral blood T (total and subsets) and NK cells.

To estimate the anti-tumor activity of ALT-803 by radiologic or pathologic disease

response, progression free survival, and overall survival in treated patients.

To characterize the immunogenicity and pharmacokinetic profile, including serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ and TNF-α, of ALT-803 in treated

patients.

**Study Design:** 

This is a Phase Ib/II, open-label, multi-center, competitive enrollment and dose-escalation study of ALT-803 in patients with relapsed or refractory multiple myeloma.

The study includes a dose escalation phase to determine the MTD or MED using a modified classic (3+3) dose escalation design and to designate a dose level for the Phase II expansion phase (RP2D) and a two-stage expansion phase at the RP2D using a Simon two-stage design. In Phase I, five dose levels will be evaluated. A step-down dose level (cohort# -1) will be provided in the event of encountering DLT in two patients at the planned initial dose level. In the absence of unacceptable toxicity or disease progression, each enrolled patient will receive up to four 6-week study treatment cycles, each consisting of a 4-week treatment period and a 2-week rest period. In each cycle, patients will receive four doses of ALT-803 by intravenous injection weekly for 4 weeks followed by a 2-week rest period. Patients with sufficient recovery of toxicities from the previous treatment cycles will be eligible to continue study treatment. After receiving two treatment cycles, patients who have at least stable disease assessed at week 11-12 may receive up to two additional study treatment cycles followed by reassessment for continued tumor response.

The study will be conducted in conformity with Good Clinical Practice (GCP).

### **Treatments:**

The study treatment plan for each enrolled patient includes up to four 6-week study treatment cycles. In each cycle, patients will receive four weekly doses of ALT-803 by intravenous injection followed by a 20-day rest period. The rest period may be extended to include up to four additional weeks if necessary. Patients who do not experience or who sufficiently recover from toxicities of the previous treatment cycles will be eligible to continue the treatment included in the study treatment plan.

Treated patients will have up to two anti-tumor evaluation visits. Patients who receive at least three study drug doses during the first 2-cycle treatment period will be evaluated for anti-tumor response during week 11-12. Patients who have at least stable disease from the first anti-tumor evaluation and who meet other criteria to continue study treatment will receive up to two additional study treatment cycles, with the same treatment schedule and at the same dose level as the first two cycles, followed by reassessment for continued tumor response.

The study treatment and response evaluation schedule is illustrated below:

| Treatment Cycle | | Сус | le #1 | | REST | | Сус | le #2 | | Response<br>Evaluation | | Cyc | le #3 | | REST | ( | Cycle | | Response<br>Evaluation | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Week | Treatment Week 1 2 3 4 5-6 | | | | 5-6 | 7 | 8 | 9 | 10 | 11-12 | 13 | 14 | 15 | 16 | 17-18 | 19 | 20 | 21 | 22 | 23-24 |
| Treatment Day | reatment Day 1 8 15 22 | | 22 | 22 23-42 43 50 5 | | 57 | 64 | 65-84 | 85 | 92 | 99 | 106 | 107-126 | 127 | 134 | 141 | 148 | 149-168 | | |
| Dose# | 1 | 2 | 3 | 4 | | 5 | 6 | 7 | 8 | | 9 | 10 | 11 | 12 | | 13 | 14 | 15 | 16 | |
| Response Evaluation | | | | | Rest<br>weeks | | | | | X | | | | | Rest<br>weeks | | | | | X |
| ALT-803 | | X | X | X | | X | X | X | X | | X | X | X | X | | X | X | X | X | |

There are no restrictions on further therapies, such as chemotherapy, radiation therapy or surgery to be used after the protocol-specified therapy. Clearly, post-study treatments could be of significant clinical benefit in selected patients, and these patients will be followed for outcome.

Enrolled patients will receive the study treatment at qualified cancer treatment centers with adequate diagnostic and treatment facilities to provide appropriate management of therapy and complications. ALT-803 will be administered by intravenous infusion into a central or peripheral vein under the supervision of a qualified physician experienced in the use of biologic anti-cancer agents.

# **Dose Escalation Phase:**

A modified 3 + 3 design will be used for identifying a tolerable dose for phase II studies by monitoring patients for DLTs to determine the MTD and for identifying an efficacious dose by monitoring patients' ALC and WBC count to determine the MED during the DLT observation period. The dose escalation phase is concluded when either the MTD or the MED is determined. A dose level (RP2D) will then be designated for Phase II study. There are five escalating dose levels of ALT-803 and a step-down cohort (-1) with a lower dose level of ALT-803 in the event that unexpected toxicity is encountered at the initial dose level.

Below are the planned dose levels of the study drug during the dose escalation phase of the study.

| Cohort | ALT-803 Dose (µg/kg) | Number of patients |
|-------------|----------------------|--------------------|
| -1 | 0.5 | 3 to 6 |
| 1 (initial) | 1 | 3 to 6 |
| 2 | 3 | 3 to 6 |
| 3 | 6 | 3 to 6 |
| 4 | 10 | 3 to 6 |
| 5 | 20 | 3 to 6 |

Dose limiting toxicity (DLT) is defined as follows: any toxicity that is not clearly unrelated to drug administration that is of Grade 3 and does not resolve to Grade 1 or lower within a week despite the use of medical intervention or that is of Grade 4, with exceptions described in the study protocol.

The DLT Observation Period is defined as the duration of the first treatment cycle.

Maximum Tolerated Dose level (MTD) is defined as a dose level at which <2 out of 6 patients experienced DLT and that is one level below a dose that was not tolerated.

Minimal Efficacious Dose (MED) is defined as a dose level which produces an ALC  $\geq$ 25,000/µL sustained for 14 days or a total WBC  $\geq$ 35,000/µL sustained for 14 days among 2/3 or 4/6 of patients. For safety, we have also defined an "exceeding MED" as the occurrence of ALC  $\geq$ 35,000/µL or WBC  $\geq$ 50,000/µL sustained for 14 days.

# **Expansion Phase**

The two-stage expansion phase at the MTD or the MED level will be conducted using an optimal Simon's two-stage design. Objective response (OR) (defined as complete response (CR) + partial response (PR)) will be evaluated and set thresholds of lack of efficacy (OR rate (ORR) = 10%) and an efficacy level of interest (ORR = 30%) will be selected.

### **Stopping Rules:**

Patient enrollment will be temporarily suspended based on occurrence of any of the following events, and the study committee, including the sponsor, the Data Safety Monitoring Board and principal investigators will meet to discuss how to proceed with future patient enrollment in the study.

During the dose escalation phase of the study,

• If the maximum planned dose level has been reached, but neither the MTD nor MED can be determined.

• If de-escalation occurs and the step-down dose level cannot be designated as the MTD or MED.

Any time during the expansion phase of the study,

- More than 33% of patients experience a possible, probable or definite study drug related DLT.
- Favorable anti-tumor response data collected from enrolled patients.

At any time during the study,

The study committee may meet to discuss how to proceed with the study and may make any or all of the following recommendations for further patient enrollment:

- Downward adjust the study drug dose.
- Adjust the study drug dosing schedule.
- Recommend more effective pre-therapy, intra-therapy and post-therapy side effect mitigation interventions.
- Correct protocol technical errors that caused unnecessary dose omissions or premature treatment discontinuations. After correction of protocol errors, the DSMB may meet to re-evaluate the safety profile of the study treatment and recommend how to proceed with the study, if necessary.

#### **Evaluations:**

Patients will be evaluated for clinical toxicities during the treatment. Patients' blood samples will be collected to assess the pharmacokinetic profile and immunogenicity of the study drug. The anti-tumor response will be evaluated at week 11-12 and week 23-24 from the start of study treatment. All patients who receive at least 3 doses of the study drug ALT-803 will be included in the anti-tumor response evaluation.

### Population:

Patients of 18 years of age and above with relapsed or refractory multiple myeloma. Patients also need to have adequate cardiac, pulmonary, liver and kidney functions and have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

### **Sample Size:**

A total of up to 30 assessable patients will be accrued to the dose escalation phase of the study (Phase Ib). Anticipated enrollment to this phase is 18 patients. Up to an additional 23 assessable patients will be enrolled at the expansion phase (Stage 1 and 2) of the study (Phase II). A total of approximately 41 assessable patients will be enrolled to complete the study. Assuming a 20% rate of ineligible or non-assessable cases, a total of up to 50 patients may be accrued to the study.

# Primary Endpoints

For Phase Ib only

(1) Determination of the MTD or MED and designation of the recommended dose level (RP2D) for Phase II study of ALT-803 in patients with relapsed or refractory multiple myeloma.

### For Phase Ib & II

- (2) Safety profile of ALT-803 in treated patients.
- (3) Disease response rate of treated patients.

### **Secondary**

### **Endpoints**

- (1) Evaluation of the effect of ALT-803 on the peripheral ALC and WBC counts, the number and phenotype of peripheral blood T (total and subsets) and NK cells in treated patients.
- (2) Duration of response in treated patients.
- (3) Progression free survival of treated patients.
- (4) Overall survival of treated patients.
- (5) Characterization of the immunogenicity and pharmacokinetic profile, including serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ and TNF-α, of ALT-803 in treated patients.

## Pharmacokinetics & Biomarkers:

Fresh blood samples will be collected to assess immune cell levels and phenotype, and serum samples for pharmacokinetics, immunogenicity of the study drug ALT-803, and the serum levels of IL-2, IL-4, IL-6, IL-10, IFN- $\gamma$  and TNF- $\alpha$  after ALT-803 administration in treated patients. Blood samples for pharmacokinetic analysis will be taken on the first day of ALT-803 administration in the first study treatment cycle. Venous blood will be obtained at Time 0 (before the start of infusion), at 30 minutes, and 2, 4, 6 and 24 hours from Time 0 for the assessment of ALT-803 serum concentrations. Non-compartmental and compartmental analyses will be conducted. In addition, the same blood samples collected for PK analysis will be used to assess the serum levels of IL-2, IL-4, IL-6, IL-10, IFN- $\gamma$  and TNF- $\alpha$ . Fresh blood samples for immune cell levels and phenotype testing will be collected before the start of first and fourth dose of study drug infusion in each treatment cycle. Bone marrow samples will be collected for future analysis of molecular markers associated with responses or resistance to ALT-803 in patients with relapsed or refractory multiple myeloma.

### **Monitoring Tests:**

Blood samples for standard chemistry and CBC with differential will be obtained at screening, on each study drug infusion day, and at follow-up visits. Blood samples for immunogenicity testing for anti-ALT-803 antibodies will be collected prior to dosing on the first ALT-803 infusion day and at weeks 7 and 12 from the initial dose of study treatment. Blood and urine samples will be collected on each follow-up visit for response assessment.

## Response Assessment:

There are at least two response assessments for treated patients: the first assessment during week 11-12 and the second assessment during week 23-24 from the start of study treatment. After completion of the first two cycles of study treatment, patients who have received at least 3 doses of study drug will have the first response assessment. After completion of the two additional cycles of study treatment, patients, regardless of the number of additional study drug doses received, will have the second response assessment. Response assessments will be carried out according to the new International Uniform Response Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. Baseline evaluations should be performed up to 14 days before study treatment starts.

# Progression & Survival

#### **Assessment:**

Progression-free survival, overall survival, and duration of response of all treated patients will be assessed every three months during year 1 and then every 6 months during years 2 and 3 from the start of study treatment, or through the point designated as the end of the study follow up.

#### **Adverse Events:**

All patients will be monitored and evaluated for clinical toxicities during the treatment period and queried at each follow-up visit for Adverse Events (AEs). Patients may volunteer information concerning AEs. All adverse events will be graded by using the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0), and logged in the patient Case Report Form. The study centers should report all Serious Adverse Events (SAEs) and all events that trigger patient's study treatment discontinuation to the sponsor via phone, fax or email (or a combination) no more than 24 hours after learning of the event. The sponsor will use the information to manage and coordinate the dose escalation, cohort expansion and patient enrollment. The sponsor will then inform all of the participating clinical sites of the current dose level and the number of patients to be enrolled at that level, or of any patient enrollment suspension via phone, fax or email within 24 hours of learning of the event. The study centers should report all other adverse events to the sponsor following the guidelines defined in the study protocol. All study drug related AEs that are both serious and unexpected will be reported to the FDA in an expedited manner in accordance with 21 CFR §312.32.

### **Statistical Plan:**

For each cohort, all AEs will be tabulated and examined and all safety, pharmacokinetic and tumor response data will be evaluated. For estimation of duration of response and progression free survival, the Kaplan-Meier method will be used. P-values of  $\leq 0.05$  (two-sided) will be considered to indicate statistical significance.

### 8. STUDY CALENDAR, CLINICAL PROCEDURES & TESTS

### 8.1 Study calendar

| TESTS & PROCEDURES | SCREEN/<br>BASELINE <sup>1</sup> | | REAT | | | REST | | REAT! | | Γ | 1 <sup>ST</sup> RESPONSE<br>ASSESSMENT | TREATMENT CYCLES #3 AND #4 | 2 <sup>ND</sup> RESPONSE<br>ASSESSMENT | FOLLOW-UPS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | | | | 1 | | | | 2<br>7 8 9 10 | | 3 | 4-5 | 6 | 9 12 18 24 30 36 | |
| Study Week | | 1 | 2 | 3 | 4 | 5-6 | 7 | | | 11-12 | 13-22 | 23-24 | | |
| Study Day | | 1 | 8 | 15 | 22 | 23-42 | 43 | 50 | 57 | 64 | 65-84 | 85-148 | 149-168 | Any day during the month |
| Tolerance Window | | | +/- 2 | days | | 23-42 | | +/- 2 0 | days | | Any day | | Any day | |
| Medical history | X | | | | | | | | | | | | | |
| Serum pregnancy test <sup>2</sup> | X | | | | | | | | | | | Follow Institution's | | |
| Complete physical exam | X | X | | | | | X | | | | X | standard of care (SOC) | X | |
| Vital signs, Weight, Height <sup>3</sup> , Cardiac & Lung function monitoring | X | X | X | X | X | | X | X | X | X | X | policy. If performed, follow the | X | |
| Concurrent medication | X | X | X | X | X | | X | X | X | X | X | same schedule as in the | X | |
| Adverse event assessment <sup>4</sup> | X | X | X | X | X | | X | X | X | X | X | first two cycles of study | X | |
| CBC with Differential | X | X | X | X | X | R | X | X | X | X | X | treatment. | X | |
| Blood Chemistry | X | X | X | X | X | E | X | X | X | X | X | | X | |
| EKG | X | $X^5$ | | | | | X | | | | | | | |
| PFT only when clinically indicated | X | | | | | S | | | | | | | | |
| Response evaluation <sup>6</sup> | | | | | | Т | | | | | X | | X | |
| Serum quantitative immunoglobulins | X | | | | | | | | | | X | | X | |
| SPEP | X | | | | | P | | | | | X | | X | |
| UPEP-random | X | | | | | • | | | | | X | | X | |
| SIFE | X | | | | | E | | | | | X | | X | |
| UIFE -random | X | | | | | R | | | | | X | | X | |
| Serum FLC assay <sup>6.1</sup> | X | | | | | | | | | | X | | X | |
| Bone marrow plasma cell percentage <sup>6.2</sup> | X | | | | | I | | | | | X | | X | |
| Bone marrow immunohistochemistry or immunofluorescence <sup>6,3</sup> | | | | | | О | | | | | X | | X | |
| Soft tissue plasmacytomas assessment <sup>6.4</sup> | | | | | | R | | | | | X | | X | |
| Disease & survival follow-up/post-therapies <sup>7</sup> | | | | | | | | | | | | | | X X X X X X |
| Immune cell levels & phenotype <sup>8,11</sup> | | $X^8$ | | | $X^8$ | | $X^8$ | | | $X^8$ | | | | |
| PK <sup>x</sup> , IL-2, IL-4, IL-6, IL-10, IFN-γ, TNF-α <sup>9,11</sup> | | $X^9$ | | | İ | | | | | | | | | |
| Immunogenicity tests <sup>10, 11</sup> | | $X^{10}$ | | | | | X | X | | X | | | | |
| Study drug (ALT-803) | | a1 | a2 | a3 | a4 | | a5 | a6 | a7 | a8 | | Follow the same schedule as in the first 2 cycles of study treatment | | |

Screening/baseline evaluations are performed ≤ 14 days prior to start of therapy. If the patient's condition is deteriorating, ECOG status and laboratory evaluations should be repeated within 48 hours initiation of study treatment infusion. Pregnancy test is for women with childbearing potential only. Vital signs (especially blood pressure), clinical status and laboratory tests should be reviewed before start of therapy. Vital signs will be evaluated at 15, 30, 60 and 120 minutes and then hourly post infusion until discharge (or at completion of dose monitoring) from the clinic, and body weight before infusion on drug infusion day. Patients who have an on-going study drug-related SAE upon study completion or at discontinuation of study will be contacted by the investigator or his/her designee every week until the event is resolved or determined to be irreversible. If the screening EKG was performed within 14 days prior to start of study treatment, the EKG is not required. Bisease response and progression assessment will be evaluated using the new International Uniform Response Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. Uniform Desponse Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. Uniform Serum and urine M-protein are unmeasurable and bone marrow plasma cell percentage > 30% at baseline. Only when scra is to be determined. Only when present at baseline, and to confirm CR or PR by X-rays, MRI or CT scans. Information about tumor assessment & other therapies received after completion of study treatment will be collected if available. Fresh blood samples for immune cell levels & phenotype testing will be collected before dosing. Collect blood samples at Time 0 (before drug infusion), at 30 min (+/- 5 min), 2 hour (+/- 15 min), 4 hour (+/- 30 min), 6 hour (+/- 60 min), 24 hour (+/- 60 min), 24 hour (+/- 60 min), 24 hour (+/- 60 min), 24 hour (+/- 60 min), 25 hour (+/- 60 min), 25 hour (+/- 60 min), 25 hour (+/- 60 min), 25 hour (+/- 60 mi

### CLINICAL STUDY PROTOCOL

CA-ALT-803-02-13 **Protocol Number:** 

A Study of ALT-803 in Patients with Relapsed or Refractory Multiple Myeloma **Protocol Title:** 

**Date of Protocol:** 

January 7, 2014 Version# 01 Version# 02 February 3, 2014 Version# 03 February 5, 2014

**Sponsor Contact:** Altor BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

## **Table of Contents**

| 2 | YNOPSI | | 6 |
|---|---|---|---|
| 1. | OBJ | ECTIVES | 12 |
| | 1.1 | Primary objectives | 12 |
| | 1.2 | SECONDARY OBJECTIVES | |
| 2. | | KGROUND | |
| | 2.1 | ALT-803 – General information | |
| | 2.2 | MULTIPLE MYELOMA | |
| | 2.3 | IMMUNE-BASED THERAPIES FOR CANCER | |
| | 2.4 | PHARMACOLOGICAL EFFECTS OF ALT-803 IN VITRO AND IN ANIMALS | |
| | 2.4.1 | Development of ALT-803 (IL-15N72D:IL-15RaSu/IgG1 Fc complex) | |
| | 2.4.2 | | |
| | 2.4.3 | | |
| | 2.4.4 | | |
| | 2.4.5 | | |
| | 2.5 | NON-CLINICAL TOXICOLOGY | 17 |
| | 2.5.1 | Multi-dose toxicity studies in mice | 17 |
| | 2.5.2 | | |
| | 2.6 | PHARMACOKINETICS | |
| | 2.6.1 | | |
| | 2.6.2 | 1 | |
| | 2.7 | RATIONALE FOR HUMAN CLINICAL STARTING DOSE | |
| | 2.8 | HUMAN EXPERIENCE | 20 |
| 3. | RAT | TIONALE FOR THE CURRENT STUDY | 21 |
| 4. | OVE | ERALL STUDY DESIGN | 22 |
| 5. | | DY POPULATION | |
| ٥. | 5.1 | INCLUSION CRITERIA | |
| | 5.2 | EXCLUSION CRITERIA. | |
| | 5.3 | INCLUSION OF WOMEN AND MINORITIES | |
| , | | | |
| 6. | | DY DESIGN | |
| | 6.1 | STUDY FLOW DIAGRAM | |
| | 6.2 | SCREENING AND ENROLLMENT | |
| | 6.3 | STUDY TREATMENT | |
| | 6.3.1 | | |
| | 6.3.2 | | |
| | 6.3.3 | V 01 1 | |
| | 6.3.4<br>6.3.5 | 7 | |
| | 6.4 | Pre and post-therapy intervention guidelines DURATION OF PATIENT PARTICIPATION | |
| | 6.5 | DOSE ESCALATION PHASE | |
| | 6.6 | | |
| | | EXPANSION PHASE | |
| | 6.7 | STOPPING RULES | |
| | 6.7.1<br>6.7.2 | | |
| | 6.7.3 | At any time during the study | |
| | 6.8 | PATIENT MONITORING, RESPONSE EVALUATION, DISEASE PROGRESSION & SURVIVAL FOLLOW-UP | |
| | 6.8.1 | Patient monitoring | |
| | 6.8.2 | Response evaluation. | |
| | 6.8.3 | | |

| | 6.9 I | OSE LIMITING TOXICITY | 32 |
|---|---|---|---|
| | 6.9.1 | Definition of dose limiting toxicity | |
| | 6.9.2 | Definition of maximum tolerated dose (MTD) | |
| | 6.9.3 | Definition of minimal efficacious dose (MED) | |
| | 6.10 | STUDY TREATMENT DISCONTINUATION | 33 |
| | 6.10.1 | Study treatment discontinuation events | 3. |
| | 6.10.2 | Replacement of participants | 3. |
| | 6.10.3 | Follow-ups after treatment discontinuation | 3. |
| | 6.10 | 0.3.1. Discontinuation due to SAEs or on-going study drug related AEs | |
| | 6.10 | 0.3.2. Discontinuation due to any other reasons | 3: |
| | 6.11 | STUDY TREATMENT INTERRUPTION | 35 |
| | 6.11.1 | Kidney dysfunction | |
| | 6.11.2 | Hematological dysfunction | |
| | 6.11.3 | Hypotension | |
| | 6.11.4 | Allergic reactions and cytokine release syndrome/acute infusion reaction | |
| | 6.12 | GENERAL SUPPORTIVE CARE GUIDELINES AND DRUG INTERACTION | |
| | 6.12.1 | Hypotension and capillary leak syndrome | |
| | 6.12.2 | Pulmonary dysfunction | |
| | 6.12.3 | Impaired kidney and liver functions | |
| | 6.12.4 | Infection | |
| | 6.12.5 | Fever and chills | |
| | 6.12.6 | Gastritis | |
| | 6.12.7 | Diarrhea, nausea and vomiting | |
| | 6.12.8 | Pruritus and dermatitis | |
| | 6.12.9 | Acidosis | |
| | 6.12.1 | | |
| | 6.12.1 | | |
| | 6.12.1. | | |
| | | e e e e e e e e e e e e e e e e e e e | |
| 7 | STU | V DRUG: AVAILABILITY ACCOUNTABILITY PACKAGING & LARFLING | 30 |
| 7. | | OY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | |
| | 7.1 | AVAILABILITY | 39 |
| | 7.1 <i>I</i> 7.2 <i>I</i> 7.2 | AVAILABILITY | 39 |
| | 7.1 7.2 7.3 I | AVAILABILITY<br>ACCOUNTABILITY<br>PACKAGING | 39 |
| | 7.1 7.2 7.3 I | AVAILABILITY | 39 |
| | 7.1 7.2 7.3 1.7.4 1.1 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING | 39<br>39<br>39 |
| 8. | 7.1 A<br>7.2 A<br>7.3 I<br>7.4 I | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING OY CALENDAR, CLINICAL PROCEDURES & TESTS | 39<br>39<br>39 |
| 8. | 7.1 2<br>7.2 2<br>7.3 1<br>7.4 1<br>STUE<br>8.1 5 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING OY CALENDAR, CLINICAL PROCEDURES & TESTS | 39<br>39<br>39<br>40 |
| 8. | 7.1 7.2 7.3 1.7.4 1.7.4 1.5 STUE 8.1 5.8.2 1.5 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING CALENDAR, CLINICAL PROCEDURES & TESTS CTUDY CALENDAR PROCEDURE AND TESTS | 39<br>39<br>39<br>40 |
| 8. | 7.1 7.2 7.3 1.7.4 1.7.4 1.5 STUE 8.1 8.2 1.8.2.1 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING OY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype | 39<br>39<br>39<br>40<br>40 |
| 8. | 7.1 7.2 7.3 1.7.4 1.7.4 1.5 STUE 8.1 8.2 1.8.2.1 8.2.2 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING OY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy | 39<br>39<br>39<br>40<br>41 |
| 8. | 7.1 7.2 7.3 1.7.4 1.5 STUE 8.1 8.2 1.8.2.2 8.2.3 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING LABELING OY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test | 39<br>39<br>40<br>41<br>44<br>44 |
| 8. | 7.1 7.2 7.3 1.7.4 1.5 STUE 8.1 8.2.1 8.2.2 8.2.3 8.2.4 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING OY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test. Physical examination | 39<br>39<br>39<br>40<br>4<br>4<br>4 |
| 8. | 7.1 7.2 7.3 1.7.4 1.5 STUE 8.1 8.2 1.8.2.2 8.2.3 8.2.4 8.2.5 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING LABELING DY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height | 39<br>39<br>39<br>40<br>4<br>4<br>4<br>4<br>4 |
| 8. | 7.1 7.2 7.3 1.7.4 1.5 STUE 8.1 8.2 1.8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING BY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment | 39<br>39<br>39<br>40<br>4<br>4<br>4<br>4<br>4<br>4 |
| 8. | 7.1 7.2 7.3 1.7.4 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING LABELING OY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring | 39<br>39<br>40<br>4 |
| 8. | 7.1 7.2 7.3 1.7.4 | AVAILABILITY ACCOUNTABILITY PACKAGING ABELING DY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring Clinical blood tests | 39<br>39<br>40<br>4 |
| 8. | 7.1 7.2 7.3 1.7.4 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING DY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring Clinical blood tests Disease assessment tests and procedures | 39<br>39<br>40<br>44 |
| 8. | 7.1 7.2 7.3 1.7.4 1.7.4 1.7.4 1.7.4 1.7.5 STUE 8.1 8.2.1 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 8.2.8 8.2.9 8.2.10 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING PY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring Clinical blood tests Disease assessment tests and procedures Adverse event assessment | 39<br>39<br>39<br>40<br>4 |
| 8. | 7.1 7.2 7.3 1.7.4 1.7.4 1.7.4 1.7.4 1.7.5 STUE 8.1 8.2.1 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 8.2.8 8.2.9 8.2.10 8.2.11 | AVAILABILITY ACCOUNTABILITY PACKAGING LABELING PY CALENDAR, CLINICAL PROCEDURES & TESTS STUDY CALENDAR PROCEDURE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test. Physical examination Vital signs, body weight & height Cardiac assessment Pulmonary function monitoring Clinical blood tests Disease assessment tests and procedures Adverse event assessment Response assessment | 39<br>39<br>39<br>40<br>4 |
| 8. | 7.1 7.2 7.3 1.7.4 1.5 STUE 8.1 8.2.1 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 8.2.8 8.2.9 8.2.10 8.2.11 8.2.12 | AVAILABILITY | 39<br>39<br>39<br>40<br>40<br>4 |
| 8. | 7.1 7.2 7.3 1.7.4 1.5 STUE 8.1 8.2.1 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 8.2.8 8.2.9 8.2.10 8.2.11 8.2.12 8.2.13 | AVAILABILITY ACCOUNTABILITY ACCOUNTA | 39<br>39<br>39<br>40<br>40<br>4 |
| 8. | 7.1 7.2 7.3 1.7.4 1.7.4 1.7.4 1.7.4 1.7.4 1.7.5 STUE 8.1 8.2.1 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 8.2.8 8.2.9 8.2.11 8.2.12 8.2.13 8.2.14 | AVAILABILITY ACCOUNTABILITY ACCOUNTA | 39<br>39<br>39<br>40<br>40<br>4 |
| 8. | 7.1 7.2 7.3 1.7.4 1.7.4 1.7.4 1.7.4 1.7.4 1.7.5 STUE 8.1 8.2.1 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 8.2.8 8.2.9 8.2.10 8.2.11 8.2.12 8.2.13 8.2.14 8.2.15 | AVAILABILITY ACCOUNTABILITY ACCOUNTABILITY ACCOUNTABILITY ACCOUNTABILITY ACCOUNTABILITY ACCOUNTABILITY ABELING ABELING ASELING ASELING ASELING ASTORY ASSAYS (CONTINUATE AND TESTS Assays for immune cell levels and phenotype Medical history & prior therapy Pregnancy test. Physical examination Vital signs, body weight & height Cardiac assessment. Pulmonary function monitoring Clinical blood tests Disease assessment tests and procedures Adverse event assessment Response assessment Disease progression and survival follow-up Pharmacokinetic (PK) testing Biomarker assays for IL-2, IL-4, IL-6, IL-10, IFN-\gamma and TNF-\alpha Immunogenicity tests - detection of anti-ALT-803 antibodies | 39<br>39<br>39<br>40<br>40<br>41<br>42<br>44 |
| 8. | 7.1 7.2 7.3 1.7.4 1.7.4 1.7.4 1.7.4 1.7.4 1.7.5 STUE 8.1 8.2.1 8.2.2 8.2.3 8.2.4 8.2.5 8.2.6 8.2.7 8.2.8 8.2.9 8.2.10 8.2.11 8.2.12 8.2.13 8.2.14 8.2.15 | AVAILABILITY ACCOUNTABILITY ACCOUNTA | 39<br>39<br>39<br>40<br>40<br>41<br>42<br>44 |

| 9.2 EFFECT ASSESSMENT SCHEDULE | 44 |
|-----------------------------------------------------------------|----|
| 9.3 METHODOLOGY OF RESPONSE EVALUATION | 44 |
| 9.4 RESPONSE EVALUATION CRITERIA | 45 |
| 9.5 DISEASE PROGRESSION EVALUATION CRITERIA | 46 |
| 10. STATISTICAL ANALYSIS | 47 |
| 10.1 Study objectives | 47 |
| 10.2 Sample size | 47 |
| 10.3 DATA COLLECTION | |
| 10.4 Data analysis | 47 |
| 10.4.1 Analysis of safety | 48 |
| 10.4.2 Analysis of response | |
| 10.4.3 Pharmacokinetics | 48 |
| 11. REGULATORY AND REPORTING REQUIREMENTS | 49 |
| 11.1 ADVERSE EVENTS RECORDING, REPORTING AND COMMUNICATION | |
| 11.2 ADVERSE EVENT TERMINOLOGY AND DEFINITIONS | |
| 11.3 ADVERSE EVENT REPORTING PROCEDURES | |
| 11.4 ADVERSE EVENT EXPEDITED REPORTING GUIDELINES | |
| 11.5 SUBMISSION OF SERIOUS ADVERSE EVENT REPORTING | |
| 11.6 Data Reporting Forms | |
| 11.7 REPORT /DATA SUBMISSION ADDRESS & CONTACT | |
| 11.8 PATIENT RECORDS, QUALITY ASSURANCE, RECORDS RETENTION | |
| 11.9 Method of review | |
| 11.10 SPECIAL REGULATORY CONSIDERATIONS | |
| 11.10.1 HIPAA | |
| 11.10.2 Protocol amendments, informed consent, and IRB approval | |
| 12. CONFIDENTIALITY | |
| 13. ETHICAL STANDARDS & INVESTIGATOR OBLIGATIONS | 53 |
| 14. LIST OF EXPECTED ADVERSE EVENTS | 54 |
| 15. CTCAE | 56 |
| REFERENCES | 57 |
| APPENDIX A: ECOG | |
| APPENDIX B: NEW YORK HEART ASSOCIATION CLASSIFICATION | |
| APPENDIX C: ETHICAL STANDARDS | |
| APPENDIX D: INVESTIGATOR OBLIGATIONS | |
| APPENDIX E: CONTACT LIST - ALTOR | |
| APPENDIX F: CONTACT LIST – DATA SAFETY MONITORING BOARD (DSMB) | |
| APPENDIX G: CONTACT LIST - LABORATORIES | 66 |

#### **SYNOPSIS**

**Sponsor:** Altor Bioscience Corporation

**Protocol#:** CA-ALT-803-02-13

Study Drug Name: Not applicable

**Study Treatment** 

Active agents: ALT-803, a "recombinant human super agonist interleukin-15 (IL-15) complex"

(AKA, IL-15N72D:IL-15RαSu/IgG1 Fc complex)

**Study Type:** Interventional

Study Phase: Ib/II

**Protocol Title:** A Study of ALT-803 in Patients with Relapsed or Refractory Multiple Myeloma

**Objectives:** To evaluate the safety and tolerability of escalating doses, identify the Maximum Tolerated Dose level (MTD) or Minimum Efficacious Dose (MED) and designate

a dose level for Phase II study (RP2D) of ALT-803 in patients with relapsed or

refractory multiple myeloma.

To evaluate the effect of ALT-803 on the peripheral absolute lymphocyte counts (ALC) and white blood cell (WBC) counts, the number and phenotype of

peripheral blood T (total and subsets) and NK cells.

To estimate the anti-tumor activity of ALT-803 by radiologic or pathologic disease

response, progression free survival, and overall survival in treated patients.

To characterize the immunogenicity and pharmacokinetic profile, including serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ and TNF-α, of ALT-803 in treated

patients.

**Study Design:** 

This is a Phase Ib/II, open-label, multi-center, competitive enrollment and dose-escalation study of ALT-803 in patients with relapsed or refractory multiple myeloma.

The study includes a dose escalation phase to determine the MTD or MED using a modified classic (3+3) dose escalation design and to designate a dose level for the Phase II expansion phase (RP2D) and a two-stage expansion phase at the RP2D using a Simon two-stage design. In Phase I, five dose levels will be evaluated. A step-down dose level (cohort# -1) will be provided in the event of encountering DLT in two patients at the planned initial dose level. In the absence of unacceptable toxicity or disease progression, each enrolled patient will receive up to four 6-week study treatment cycles, each consisting of a 4-week treatment period and a 2-week rest period. In each cycle, patients will receive four doses of ALT-803 by intravenous injection weekly for 4 weeks followed by a 2-week rest period. Patients with sufficient recovery of toxicities from the previous treatment cycles will be eligible to continue study treatment. After receiving two treatment cycles, patients who have at least stable disease assessed at week 11-12 may receive up to two additional study treatment cycles followed by reassessment for continued tumor response.

The study will be conducted in conformity with Good Clinical Practice (GCP).

### **Treatments:**

The study treatment plan for each enrolled patient includes up to four 6-week study treatment cycles. In each cycle, patients will receive four weekly doses of ALT-803 by intravenous injection followed by a 20-day rest period. The rest period may be extended to include up to four additional weeks if necessary. Patients who do not experience or who sufficiently recover from toxicities of the previous treatment cycles will be eligible to continue the treatment included in the study treatment plan.

Treated patients will have up to two anti-tumor evaluation visits. Patients who receive at least three study drug doses during the first 2-cycle treatment period will be evaluated for anti-tumor response during week 11-12. Patients who have at least stable disease from the first anti-tumor evaluation and who meet other criteria to continue study treatment will receive up to two additional study treatment cycles, with the same treatment schedule and at the same dose level as the first two cycles, followed by reassessment for continued tumor response.

The study treatment and response evaluation schedule is illustrated below:

| Treatment Cycle | | Сус | le #1 | | REST Cycle # | | | | | Response<br>Evaluation | | Cycl | le #3 | | REST | Cycle #4 | | | | Response<br>Evaluation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Week | 1 | 2 | 3 | 4 | 5-6 | 7 | 8 | 9 | 10 | 11-12 | 13 | 14 | 15 | 16 | 17-18 | 19 | 20 | 21 | 22 | 23-24 |
| Treatment Day | 1 | 8 | 15 | 22 | 23-42 | 43 | 50 | 57 | 64 | 65-84 | 85 | 92 | 99 | 106 | 107-126 | 127 | 134 | 141 | 148 | 149-168 |
| Dose# | 1 | 2 | 3 | 4 | | 5 | 6 | 7 | 8 | | 9 | 10 | 11 | 12 | | 13 | 14 | 15 | 16 | |
| Response Evaluation | | | | | Rest<br>weeks | | | | | X | | | | | Rest<br>weeks | | | | | X |
| ALT-803 | | X | X | X | | X | X | X | X | | X | X | X | X | | X | X | X | X | |

There are no restrictions on further therapies, such as chemotherapy, radiation therapy or surgery to be used after the protocol-specified therapy. Clearly, post-study treatments could be of significant clinical benefit in selected patients, and these patients will be followed for outcome.

Enrolled patients will receive the study treatment at qualified cancer treatment centers with adequate diagnostic and treatment facilities to provide appropriate management of therapy and complications. ALT-803 will be administered by intravenous infusion into a central or peripheral vein under the supervision of a qualified physician experienced in the use of biologic anti-cancer agents.

# **Dose Escalation Phase:**

A modified 3 + 3 design will be used for identifying a tolerable dose for phase II studies by monitoring patients for DLTs to determine the MTD and for identifying an efficacious dose by monitoring patients' ALC and WBC count to determine the MED during the DLT observation period. The dose escalation phase is concluded when either the MTD or the MED is determined. A dose level (RP2D) will then be designated for Phase II study. There are five escalating dose levels of ALT-803 and a step-down cohort (-1) with a lower dose level of ALT-803 in the event that unexpected toxicity is encountered at the initial dose level.

Below are the planned dose levels of the study drug during the dose escalation phase of the study.

| Cohort | ALT-803 Dose (µg/kg) | Number of patients |
|-------------|----------------------|--------------------|
| -1 | 0.5 | 3 to 6 |
| 1 (initial) | 1 | 3 to 6 |
| 2 | 3 | 3 to 6 |
| 3 | 6 | 3 to 6 |
| 4 | 10 | 3 to 6 |
| 5 | 20 | 3 to 6 |

Dose limiting toxicity (DLT) is defined as follows: any toxicity that is not clearly unrelated to drug administration that is of Grade 3 and does not resolve to Grade 1 or lower within a week despite the use of medical intervention or that is of Grade 4, with exceptions described in the study protocol.

The DLT Observation Period is defined as the duration of the first treatment cycle.

Maximum Tolerated Dose level (MTD) is defined as a dose level at which <2 out of 6 patients experienced DLT and that is one level below a dose that was not tolerated.

Minimal Efficacious Dose (MED) is defined as a dose level which produces an ALC  $\geq$ 25,000/µL sustained for 14 days or a total WBC  $\geq$ 35,000/µL sustained for 14 days among 2/3 or 4/6 of patients. For safety, we have also defined an "exceeding MED" as the occurrence of ALC  $\geq$ 35,000/µL or WBC  $\geq$ 50,000/µL sustained for 14 days.

# **Expansion Phase**

The two-stage expansion phase at the MTD or the MED level will be conducted using an optimal Simon's two-stage design. Objective response (OR) (defined as complete response (CR) + partial response (PR)) will be evaluated and set thresholds of lack of efficacy (OR rate (ORR) = 10%) and an efficacy level of interest (ORR = 30%) will be selected.

### **Stopping Rules:**

Patient enrollment will be temporarily suspended based on occurrence of any of the following events, and the study committee, including the sponsor, the Data Safety Monitoring Board and principal investigators will meet to discuss how to proceed with future patient enrollment in the study.

During the dose escalation phase of the study,

• If the maximum planned dose level has been reached, but neither the MTD nor MED can be determined.

• If de-escalation occurs and the step-down dose level cannot be designated as the MTD or MED.

Any time during the expansion phase of the study,

- More than 33% of patients experience a possible, probable or definite study drug related DLT.
- Favorable anti-tumor response data collected from enrolled patients.

At any time during the study,

The study committee may meet to discuss how to proceed with the study and may make any or all of the following recommendations for further patient enrollment:

- Downward adjust the study drug dose.
- Adjust the study drug dosing schedule.
- Recommend more effective pre-therapy, intra-therapy and post-therapy side effect mitigation interventions.
- Correct protocol technical errors that caused unnecessary dose omissions or premature treatment discontinuations. After correction of protocol errors, the DSMB may meet to re-evaluate the safety profile of the study treatment and recommend how to proceed with the study, if necessary.

### **Evaluations:**

Patients will be evaluated for clinical toxicities during the treatment. Patients' blood samples will be collected to assess the pharmacokinetic profile and immunogenicity of the study drug. The anti-tumor response will be evaluated at week 11-12 and week 23-24 from the start of study treatment. All patients who receive at least 3 doses of the study drug ALT-803 will be included in the anti-tumor response evaluation.

### Population:

Patients of 18 years of age and above with relapsed or refractory multiple myeloma. Patients also need to have adequate cardiac, pulmonary, liver and kidney functions and have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

### **Sample Size:**

A total of up to 30 assessable patients will be accrued to the dose escalation phase of the study (Phase Ib). Anticipated enrollment to this phase is 18 patients. Up to an additional 23 assessable patients will be enrolled at the expansion phase (Stage 1 and 2) of the study (Phase II). A total of approximately 41 assessable patients will be enrolled to complete the study. Assuming a 20% rate of ineligible or non-assessable cases, a total of up to 50 patients may be accrued to the study.

# Primary Endpoints

For Phase Ib only

(1) Determination of the MTD or MED and designation of the recommended dose level (RP2D) for Phase II study of ALT-803 in patients with relapsed or refractory multiple myeloma.

#### For Phase Ib & II

- (2) Safety profile of ALT-803 in treated patients.
- (3) Disease response rate of treated patients.

### **Secondary**

### **Endpoints**

- (1) Evaluation of the effect of ALT-803 on the peripheral ALC and WBC counts, the number and phenotype of peripheral blood T (total and subsets) and NK cells in treated patients.
- (2) Duration of response in treated patients.
- (3) Progression free survival of treated patients.
- (4) Overall survival of treated patients.
- (5) Characterization of the immunogenicity and pharmacokinetic profile, including serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ and TNF-α, of ALT-803 in treated patients.

## Pharmacokinetics & Biomarkers:

Fresh blood samples will be collected to assess immune cell levels and phenotype, and serum samples for pharmacokinetics, immunogenicity of the study drug ALT-803, and the serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ and TNF-α after ALT-803 administration in treated patients. Blood samples for pharmacokinetic analysis will be taken on the first day of ALT-803 administration in the first study treatment cycle. Venous blood will be obtained at Time 0 (before the start of infusion), at 30 minutes, and 2, 4, 6 and 24 hours from Time 0 for the assessment of ALT-803 serum concentrations. Non-compartmental and compartmental analyses will be conducted. In addition, the same blood samples collected for PK analysis will be used to assess the serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ and TNF-α. Fresh blood samples for immune cell levels and phenotype testing will be collected before the start of first and fourth dose of study drug infusion in each treatment cycle. Bone marrow samples will be collected for future analysis of molecular markers associated with responses or resistance to ALT-803 in patients with relapsed or refractory multiple myeloma.

### **Monitoring Tests:**

Blood samples for standard chemistry and CBC with differential will be obtained at screening, on each study drug infusion day, and at follow-up visits. Blood samples for immunogenicity testing for anti-ALT-803 antibodies will be collected prior to dosing on the first ALT-803 infusion day and at weeks 7 and 12 from the initial dose of study treatment. Blood and urine samples will be collected on each follow-up visit for response assessment.

## Response Assessment:

There are at least two response assessments for treated patients: the first assessment during week 11-12 and the second assessment during week 23-24 from the start of study treatment. After completion of the first two cycles of study treatment, patients who have received at least 3 doses of study drug will have the first response assessment. After completion of the two additional cycles of study treatment, patients, regardless of the number of additional study drug doses received, will have the second response assessment. Response assessments will be carried out according to the new International Uniform Response Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. Baseline evaluations should be performed up to 14 days before study treatment starts.

# Progression & Survival

#### **Assessment:**

Progression-free survival, overall survival, and duration of response of all treated patients will be assessed every three months during year 1 and then every 6 months during years 2 and 3 from the start of study treatment, or through the point designated as the end of the study follow up.

#### **Adverse Events:**

All patients will be monitored and evaluated for clinical toxicities during the treatment period and queried at each follow-up visit for Adverse Events (AEs). Patients may volunteer information concerning AEs. All adverse events will be graded by using the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0), and logged in the patient Case Report Form. The study centers should report all Serious Adverse Events (SAEs) and all events that trigger patient's study treatment discontinuation to the sponsor via phone, fax or email (or a combination) no more than 24 hours after learning of the event. The sponsor will use the information to manage and coordinate the dose escalation, cohort expansion and patient enrollment. The sponsor will then inform all of the participating clinical sites of the current dose level and the number of patients to be enrolled at that level, or of any patient enrollment suspension via phone, fax or email within 24 hours of learning of the event. The study centers should report all other adverse events to the sponsor following the guidelines defined in the study protocol. All study drug related AEs that are both serious and unexpected will be reported to the FDA in an expedited manner in accordance with 21 CFR §312.32.

### **Statistical Plan:**

For each cohort, all AEs will be tabulated and examined and all safety, pharmacokinetic and tumor response data will be evaluated. For estimation of duration of response and progression free survival, the Kaplan-Meier method will be used. P-values of  $\leq 0.05$  (two-sided) will be considered to indicate statistical significance.

### 8. STUDY CALENDAR, CLINICAL PROCEDURES & TESTS

### 8.1 Study calendar

| TESTS & PROCEDURES | SCREEN/<br>BASELINE <sup>1</sup> | TREATMENT<br>CYCLE #1 | | | | REST | TREATMENT<br>CYCLE #2 | | | | 1 <sup>ST</sup> RESPONSE<br>ASSESSMENT | TREATMENT CYCLES<br>#3 AND #4 | 2 <sup>ND</sup> RESPONSE<br>ASSESSMENT | FOLLOW-UPS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | | 1 | | | | | 2 | | | | 3 | 4-5 | 6 | 9 12 18 24 30 36 |
| Study Week | | 1 | 2 | 3 | 4 | 5-6 | 7 | 8 | 9 | 10 | 11-12 | 13-22 | 23-24 | |
| Study Day | | 1 | 8 | 15 | 22 | 23-42 | 43 | 50 | 57 | 64 | 65-84 | 85-148 | 149-168 | Any day during the month |
| Tolerance Window | | | +/- 2 | days | 1 | 23-42 | | +/- 2 0 | lays | | Any day | | Any day | |
| Medical history | X | | | | | | | | | | | 1 | | |
| Serum pregnancy test <sup>2</sup> | X | | | | | | | | | | | Follow Institution's | | |
| Complete physical exam | X | X | | | | | X | | | | X | standard of care (SOC) | X | |
| Vital signs, Weight, Height <sup>3</sup> , Cardiac & Lung function monitoring | X | X | X | X | X | | X | X | X | X | X | policy. If performed, follow the | X | |
| Concurrent medication | X | X | X | X | X | | X | X | X | X | X | same schedule as in the | X | |
| Adverse event assessment <sup>4</sup> | X | X | X | X | X | | X | X | X | X | X | first two cycles of study | X | |
| CBC with Differential | X | X | X | X | X | R | X | X | X | X | X | treatment. | X | |
| Blood Chemistry | X | X | X | X | X | | X | X | X | X | X | | X | |
| EKG | X | $X^5$ | | | | E | X | | | | | | | |
| PFT only when clinically indicated | X | | | | | s | | | | | | | | |
| Response evaluation <sup>6</sup> | | | | | | Т | | | | | X | | X | |
| Serum quantitative immunoglobulins | X | | | | | | | | | | X | | X | |
| SPEP | X | | | | | P | | | | | X | | X | |
| UPEP-random | X | | | | | | | | | | X | | X | |
| SIFE | X | | | | | E | | | | | X | | X | |
| UIFE -random | X | | | | | R | | | | | X | | X | |
| Serum FLC assay <sup>6.1</sup> | X | | | | | | | | | | X | | X | |
| Bone marrow plasma cell percentage <sup>6.2</sup> | X | | | | | I | | | | | X | | X | |
| Bone marrow immunohistochemistry or immunofluorescence <sup>6.3</sup> | | | | | | О | | | | | X | | X | |
| Soft tissue plasmacytomas assessment <sup>6.4</sup> | | | | | | R | | | | | X | | X | |
| Disease & survival follow-up/post-therapies <sup>7</sup> | | | | | | | | | | | | | | X X X X X X |
| Immune cell levels & phenotype <sup>8,11</sup> | | $X^8$ | | | $X^8$ | | $X^8$ | | | $X^8$ | | | | * * * * * |
| PK <sup>x</sup> , IL-2, IL-4, IL-6, IL-10, IFN-γ, TNF-α <sup>9,11</sup> | | $X^9$ | | | | | | | | | | | | |
| Immunogenicity tests <sup>10, 11</sup> | | $X^{10}$ | | | | | X | | | | X | | | |
| Study drug (ALT-803) | | a1 | a2 | а3 | a4 | | a5 | a6 | a7 | a8 | | Follow the same schedule as in the first 2 cycles of study treatment | | |

Screening/baseline evaluations are performed ≤ 14 days prior to start of therapy. If the patient's condition is deteriorating, ECOG status and laboratory evaluations should be repeated within 48 hours prior to initiation of study treatment infusion. Pregnancy test is for women with childbearing potential only. Vital signs (especially blood pressure), clinical status and laboratory tests should be reviewed before start of therapy. Day 1 for the 1st patient of each cohort will have vital signs evaluated at 15, 30, 60 and 120 min then hourly for 6 hours post infusion and every 3 hours thereafter until discharge (24 hrs). Vital signs for the rest of the study visits and all visits for subsequent patients will be evaluated at 15, 30, 60 and 120 min and then hourly post infusion until discharge (or at completion of dose monitoring) from the clinic. Body weight will be collected before infusion on each drug infusion day for all patients. Patients who have an on-going study drug-related SAE upon study completion or at discontinuation of study will be contacted by the investigator or his/her designee every week until the event is resolved or determined to be irreversible. If the screening EKG was performed within 14 days prior to start of study treatment, the EKG is not required. Disease response and progression assessment will be evaluated using the new International Uniform Response Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. Only when serum and urine M-protein are unmeasurable. Valuation and urine M-protein and serum FLC are unmeasurable and bone marrow plasma cell percentage > 30% at baseline. Valuation of study when sCR is to be determined. The following the protein and serum FLC are unmeasurable and bone marrow plasma cell percentage > 30% at baseline. Valuation of study treatment will be collected in available. Fresh blood samples for immune cell levels & phenotype testing will be collected before dosing. Collect blood samples at Time 0 (before drug infusion), at 30 min (+

Page 40 of 66

### **CLINICAL STUDY PROTOCOL**

CA-ALT-803-02-13 **Protocol Number:** 

A Study of ALT-803 in Patients with Relapsed or Refractory Multiple Myeloma **Protocol Title:** 

**Date of Protocol:** 

January 7, 2014 Version# 01 Version# 02 February 3, 2014 Version# 03 February 5, 2014 Version# 04 May 16, 2014

**Sponsor Contact:** Altor BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

## **Table of Contents**

| SY | 'NOPSI | IS | 6 |
|---|---|---|---|
| 1. | OBJ | ECTIVES | 12 |
| | 1.1 | PRIMARY OBJECTIVES | |
| | 1.2 | SECONDARY OBJECTIVES | |
| 2. | | CKGROUND | |
| | 2.1 | ALT-803 – GENERAL INFORMATION | |
| | 2.2 | MULTIPLE MYELOMA | |
| | 2.3 | IMMUNE-BASED THERAPIES FOR CANCER | |
| | 2.4<br>2.4.1 | PHARMACOLOGICAL EFFECTS OF ALT-803 IN VITRO AND IN ANIMALS | |
| | 2.4.1 | | |
| | 2.4.3 | | |
| | 2.4.4 | | |
| | 2.4.5 | | |
| | | Non-clinical toxicology | |
| | 2.5.1 | Multi-dose toxicity studies in mice | 17 |
| | 2.5.2 | Multi-dose toxicity studies in cynomolgus monkeys | 18 |
| | 2.6 | PHARMACOKINETICS | |
| | 2.6.1 | 1 | |
| | 2.6.2 | 1 | |
| | 2.7 | RATIONALE FOR HUMAN CLINICAL STARTING DOSE | |
| | 2.8 | HUMAN EXPERIENCE | |
| 3. | RAT | TIONALE FOR THE CURRENT STUDY | 21 |
| 4. | OVE | ERALL STUDY DESIGN | 22 |
| 5. | | DY POPULATION | |
| | 5.1 | INCLUSION CRITERIA | |
| | 5.1 | EXCLUSION CRITERIA | |
| | 5.2 | INCLUSION OF WOMEN AND MINORITIES | |
| 6. | | DY DESIGN | |
| | 6.1 | STUDY FLOW DIAGRAM | - |
| | 6.2 | SCREENING AND ENROLLMENT | |
| | 6.3 | STUDY TREATMENT | |
| | 6.3.1 | 6 | |
| | 6.3.2 | | |
| | | Study drug preparation | |
| | 6.3.4 | 7 0 | |
| | 6.3.5<br>6.4 | 1 17 0 | |
| | 6.5 | DURATION OF PATIENT PARTICIPATION | |
| | | DOSE ESCALATION PHASE | |
| | 6.6 | EXPANSION PHASE | |
| | 6.7<br>6.7.1 | STOPPING RULES | |
| | O / I | During dose escalation phase of the study | 3 <i>I</i> |
| | 6.7.2 | During expansion phase of the study | 31 |
| | 6.7.2<br>6.7.3 | During expansion phase of the study | 31 |
| | 6.7.2<br>6.7.3<br>6.8 | During expansion phase of the study | 31<br>31<br>OGRESSION |
| | 6.7.2<br>6.7.3<br>6.8 | During expansion phase of the study | 31<br>31<br>OGRESSION<br>32 |

| 6.8.3 | Treatment cycle #3 & #4 | 32 |
|---|---|---|
| 6.8.4 | Disease progression and survival follow-up | 32 |
| 6.9 | Dose limiting toxicity | 32 |
| 6.9.1 | Definition of dose limiting toxicity | 32 |
| 6.9.2 | Definition of maximum tolerated dose (MTD) | 33 |
| 6.9.3 | Definition of minimal efficacious dose (MED) | 33 |
| 6.10 | STUDY TREATMENT DISCONTINUATION | |
| 6.10.1 | Study treatment discontinuation events | 33 |
| 6.10.2 | • | |
| 6.10.3 | | |
| 6.1 | 0.3.1. Discontinuation due to SAEs or on-going study drug related AEs | 35 |
| 6.1 | 0.3.2. Discontinuation due to any other reasons | 35 |
| 6.11 | STUDY TREATMENT INTERRUPTION | 35 |
| 6.11.1 | Kidney dysfunction | 35 |
| 6.11.2 | Hematological dysfunction | 35 |
| 6.11.3 | Hypotension | 35 |
| 6.11.4 | Allergic reactions and cytokine release syndrome/acute infusion reaction | 36 |
| 6.12 | GENERAL SUPPORTIVE CARE GUIDELINES AND DRUG INTERACTION | 36 |
| 6.12.1 | Hypotension and capillary leak syndrome | 36 |
| 6.12.2 | | |
| 6.12.3 | | |
| 6.12.4 | | |
| 6.12.5 | Fever and chills | 37 |
| 6.12.6 | Gastritis | 37 |
| 6.12.7 | Diarrhea, nausea and vomiting | 37 |
| 6.12.8 | | |
| 6.12.9 | | |
| 6.12.1 | y G | |
| 6.12.1 | Tr | |
| 6.12.1 | 2 Drug interaction | 37 |
| 7. STUI | DY DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | 39 |
| | Availability | |
| | ACCOUNTABILITY | |
| | PACKAGING | |
| | Labeling | |
| 8. STUI | DY CALENDAR, CLINICAL PROCEDURES & TESTS | 40 |
| 8.1 | STUDY CALENDAR | 40 |
| | PROCEDURE AND TESTS | |
| 8.2.1 | Assays for immune cell levels and phenotype | |
| 8.2.2 | Medical history & prior therapy | |
| 8.2.3 | Pregnancy test | |
| 8.2.4 | Physical examination | |
| 8.2.5 | Vital signs, body weight & height | |
| 8.2.6 | Cardiac assessment | |
| 8.2.7 | Pulmonary function monitoring | |
| 8.2.8 | Clinical blood tests | |
| 8.2.9 | Disease assessment tests and procedures | |
| 8.2.10 | | |
| 8.2.11 | | |
| 8.2.12 | | |
| 8.2.13 | | |
| 8.2.14 | ( ) | |
| 8.2.15 | | |
| | SUREMENT OF EFFECT | |
| 7. IVIIDA | SUMENIETTI OF EFFECT | TJ |
| 9.1 | MEASURABLE DISEASE | |
|---|---|---|
| 9.2 | EFFECT ASSESSMENT SCHEDULE | |
| 9.3 | METHODOLOGY OF RESPONSE EVALUATION | |
| 9.4 | RESPONSE EVALUATION CRITERIA | |
| 9.5 | DISEASE PROGRESSION EVALUATION CRITERIA | |
| 10. | STATISTICAL ANALYSIS | 48 |
| 10.1 | STUDY OBJECTIVES | 48 |
| 10.2 | SAMPLE SIZE | |
| 10.3 | DATA COLLECTION | |
| 10.4 | Data analysis | |
| 10.4 | | |
| 10.4 | | |
| 10.4 | | |
| | REGULATORY AND REPORTING REQUIREMENTS | |
| 11.1 | ADVERSE EVENTS RECORDING, REPORTING AND COMMUNICATION | |
| 11.2 | ADVERSE EVENT TERMINOLOGY AND DEFINITIONS | |
| 11.3 | ADVERSE EVENT REPORTING PROCEDURES | |
| 11.4 | ADVERSE EVENT EXPEDITED REPORTING GUIDELINES | _ |
| 11.5 | SUBMISSION OF SERIOUS ADVERSE EVENT REPORTING | |
| 11.6 | DATA REPORTING FORMS | |
| 11.7 | REPORT /DATA SUBMISSION ADDRESS & CONTACT | |
| 11.8 | PATIENT RECORDS, QUALITY ASSURANCE, RECORDS RETENTION | |
| 11.9<br>11.10 | | |
| _ | 10.1 HIPAA | |
| 11 | 10.1 III AA | 54 |
| | CONFIDENTIALITY | |
| | ETHICAL STANDARDS & INVESTIGATOR OBLIGATIONS | |
| | LIST OF EXPECTED ADVERSE EVENTS | |
| 15. | CTCAE | 57 |
| REFER | ENCES | 58 |
| APPEN | DIX A: ECOG | 60 |
| | DIX B: NEW YORK HEART ASSOCIATION CLASSIFICATION | |
| | DIX C: ETHICAL STANDARDS | |
| | DIX D: INVESTIGATOR OBLIGATIONS | |
| APPEN | DIX E: CONTACT LIST - ALTOR | 66 |
| APPEN | DIX F: CONTACT LIST – DATA SAFETY MONITORING BOARD (DSMB) | 67 |
| APPEN | DIX G: CONTACT LIST - LABORATORIES | 67 |

#### **SYNOPSIS**

**Sponsor:** Altor Bioscience Corporation

**Protocol#:** CA-ALT-803-02-13

Study Drug Name: Not applicable

**Study Treatment** 

Active agents: ALT-803, a "recombinant human super agonist interleukin-15 (IL-15) complex"

(AKA, IL-15N72D:IL-15RαSu/IgG1 Fc complex)

**Study Type:** Interventional

**Study Phase:** I/II

**Protocol Title:** A Study of ALT-803 in Patients with Relapsed or Refractory Multiple Myeloma

**Objectives:** To evaluate the safety and tolerability of escalating doses, identify the Maximum

Tolerated Dose level (MTD) or Minimum Efficacious Dose (MED) and designate a dose level for Phase II study (RP2D) of ALT-803 in patients with relapsed or

refractory multiple myeloma.

To evaluate the effect of ALT-803 on the peripheral absolute lymphocyte counts (ALC) and white blood cell (WBC) counts, the number and phenotype of

peripheral blood T (total and subsets) and NK cells.

To estimate the anti-tumor activity of ALT-803 by radiologic or pathologic disease

response, progression free survival, and overall survival in treated patients.

To characterize the immunogenicity and pharmacokinetic profile, including serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ and TNF-α, of ALT-803 in treated

patients.

**Study Design:** 

This is a Phase I/II, open-label, multi-center, competitive enrollment and dose-escalation study of ALT-803 in patients with relapsed or refractory multiple myeloma.

The study includes a dose escalation phase to determine the MTD or MED using a modified classic (3+3) dose escalation design and to designate a dose level for the Phase II expansion phase (RP2D) and a two-stage expansion phase at the RP2D using a Simon two-stage design. In Phase I, five dose levels will be evaluated. A step-down dose level (cohort# -1) will be provided in the event of encountering DLT in two patients at the planned initial dose level. In the absence of unacceptable toxicity or disease progression, each enrolled patient will receive up to four 6-week study treatment cycles, each consisting of a 4-week treatment period and a 2-week rest period. In each cycle, patients will receive four doses of ALT-803 by intravenous injection weekly for 4 weeks followed by a 2-week rest period. Patients with sufficient recovery of toxicities from the previous treatment cycles will be eligible to continue study treatment. After receiving two treatment cycles, patients who have at least stable disease assessed at week 11-12 may receive up to two additional study treatment cycles followed by reassessment for continued tumor response.

The study will be conducted in conformity with Good Clinical Practice (GCP).

#### **Treatments:**

The study treatment plan for each enrolled patient includes up to four 6-week study treatment cycles. In each cycle, patients will receive four weekly doses of ALT-803 by intravenous injection followed by a 2-week rest period. The rest period may be extended to include up to four additional weeks if necessary. Patients who do not experience or who sufficiently recover from toxicities of the previous treatment cycles will be eligible to continue the treatment included in the study treatment plan.

Treated patients will have up to two anti-tumor evaluation visits. Patients who receive at least three study drug doses during the first 2-cycle treatment period will be evaluated for anti-tumor response during week 11-12. Patients who have at least stable disease from the first anti-tumor evaluation and who meet other criteria to continue study treatment will receive up to two additional study treatment cycles, with the same treatment schedule and at the same dose level as the first two cycles, followed by reassessment for continued tumor response.

The study treatment and response evaluation schedule is illustrated below:

| Treatment Cycle | | Сус | le #1 | l | REST | | Сус | le #2 | | Response<br>Evaluation | | Cyc | le #3 | | REST | ( | Cycle | e #4 | | Response<br>Evaluation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Week | 1 | 2 | 3 | 4 | 5-6 | 7 | 8 | 9 | 10 | 11-12 | 13 | 14 | 15 | 16 | 17-18 | 19 | 20 | 21 | 22 | 23-24 |
| Treatment Day | 1 | 8 | 15 | 22 | 23-42 | 43 | 50 | 57 | 64 | 71-84 | 85 | 92 | 99 | 106 | 107-126 | 127 | 134 | 141 | 148 | 155-168 |
| Dose# | 1 | 2 | 3 | 4 | | 5 | 6 | 7 | 8 | | 9 | 10 | 11 | 12 | | 13 | 14 | 15 | 16 | |
| Response Evaluation | | | | | Rest<br>weeks | | | | | X | | | | | Rest<br>weeks | | | | | X |
| ALT-803 | X | X | X | X | | X | X | X | X | | X | X | X | X | | X | X | X | X | |

There are no restrictions on further therapies, such as chemotherapy, radiation therapy or surgery to be used after the protocol-specified therapy. Clearly, post-study treatments could be of significant clinical benefit in selected patients, and these patients will be followed for outcome.

Enrolled patients will receive the study treatment at qualified cancer treatment centers with adequate diagnostic and treatment facilities to provide appropriate management of therapy and complications. ALT-803 will be administered by intravenous infusion into a central or peripheral vein under the supervision of a qualified physician experienced in the use of biologic anti-cancer agents.

## **Dose Escalation Phase:**

A modified 3 + 3 design will be used for identifying a tolerable dose for phase II studies by monitoring patients for DLTs to determine the MTD and for identifying an efficacious dose by monitoring patients' ALC and WBC count to determine the MED during the DLT observation period. The dose escalation phase is concluded when either the MTD or the MED is determined. A dose level (RP2D) will then be designated for Phase II study. There are five escalating dose levels of ALT-803 and a step-down cohort (-1) with a lower dose level of ALT-803 in the event that unexpected toxicity is encountered at the initial dose level.

Below are the planned dose levels of the study drug during the dose escalation phase of the study.

| Cohort | ALT-803 Dose (µg/kg) | Number of patients |
|-------------|----------------------|--------------------|
| -1 | 0.5 | 3 to 6 |
| 1 (initial) | 1 | 3 to 6 |
| 2 | 3 | 3 to 6 |
| 3 | 6 | 3 to 6 |
| 4 | 10 | 3 to 6 |
| 5 | 20 | 3 to 6 |

Dose limiting toxicity (DLT) is defined as follows: any toxicity that is not clearly unrelated to drug administration that is of Grade 3 and does not resolve to Grade 1 or lower within a week despite the use of medical intervention or that is of Grade 4, with exceptions described in the study protocol.

The DLT Observation Period is defined as the duration of the first treatment cycle.

Maximum Tolerated Dose level (MTD) is defined as a dose level at which <2 out of 6 patients experienced DLT and that is one level below a dose that was not tolerated.

Minimal Efficacious Dose (MED) is defined as a dose level which produces an ALC  $\geq$ 25,000/µL sustained for 14 days or a total WBC  $\geq$ 35,000/µL sustained for 14 days among 2/3 or 4/6 of patients. For safety, we have also defined an "exceeding MED" as the occurrence of ALC  $\geq$ 35,000/µL or WBC  $\geq$ 50,000/µL sustained for 14 days.

# **Expansion Phase**

The two-stage expansion phase at the MTD or the MED level will be conducted using an optimal Simon's two-stage design. Objective response (OR) (defined as complete response (CR) + partial response (PR)) will be evaluated and set thresholds of lack of efficacy (OR rate (ORR) = 10%) and an efficacy level of interest (ORR = 30%) will be selected.

### **Stopping Rules:**

Patient enrollment will be temporarily suspended based on occurrence of any of the following events, and the study committee, including the sponsor, the Data Safety Monitoring Board and principal investigators will meet to discuss how to proceed with future patient enrollment in the study.

During the dose escalation phase of the study,

• If the maximum planned dose level has been reached, but neither the MTD nor MED can be determined.

• If de-escalation occurs and the step-down dose level cannot be designated as the MTD or MED.

Any time during the expansion phase of the study,

- More than 33% of patients experience a possible, probable or definite study drug related DLT.
- Favorable anti-tumor response data collected from enrolled patients.

At any time during the study,

The study committee may meet to discuss how to proceed with the study and may make any or all of the following recommendations for further patient enrollment:

- Downward adjust the study drug dose.
- Adjust the study drug dosing schedule.
- Recommend more effective pre-therapy, intra-therapy and post-therapy side effect mitigation interventions.
- Correct protocol technical errors that caused unnecessary dose omissions or premature treatment discontinuations. After correction of protocol errors, the DSMB may meet to re-evaluate the safety profile of the study treatment and recommend how to proceed with the study, if necessary.

#### **Evaluations:**

Patients will be evaluated for clinical toxicities during the treatment. Patients' blood samples will be collected to assess the pharmacokinetic profile and immunogenicity of the study drug. The anti-tumor response will be evaluated at week 11-12 and week 23-24 from the start of study treatment. All patients who receive at least 3 doses of the study drug ALT-803 will be included in the anti-tumor response evaluation.

#### **Population:**

Patients of 18 years of age and above with relapsed or refractory multiple myeloma. Patients also need to have adequate cardiac, pulmonary, liver and kidney functions and have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

#### **Sample Size:**

A total of up to 30 assessable patients will be accrued to the dose escalation phase of the study (Phase I). Anticipated enrollment to this phase is 18 patients. Up to an additional 23 assessable patients will be enrolled at the expansion phase (Stage 1 and 2) of the study (Phase II). An estimated total of approximately 41 assessable patients will be enrolled to complete the study. Assuming a 20% rate of ineligible or non-assessable cases, an estimated total of up to 50 patients may be accrued to the study.

### Primary Endpoints

#### For Phase I only

(1) Determination of the MTD or MED and designation of the recommended dose level (RP2D) for Phase II study of ALT-803 in patients with relapsed or refractory multiple myeloma.

#### For Phase I & II

- (2) Safety profile of ALT-803 in treated patients.
- (3) Disease response rate of treated patients.

# **Secondary Endpoints**

- (1) Evaluation of the effect of ALT-803 on the peripheral ALC and WBC counts, the number and phenotype of peripheral blood T (total and subsets) and NK cells in treated patients.
- (2) Duration of response in treated patients.
- (3) Progression free survival of treated patients.
- (4) Overall survival of treated patients.
- (5) Characterization of the immunogenicity and pharmacokinetic profile, including serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ and TNF-α, of ALT-803 in treated patients.

# Pharmacokinetics & Biomarkers:

Fresh blood samples will be collected to assess immune cell levels and phenotype, and serum samples for pharmacokinetics, immunogenicity of the study drug ALT-803, and the serum levels of IL-2, IL-4, IL-6, IL-10, IFN- $\gamma$  and TNF- $\alpha$  after ALT-803 administration in treated patients. Blood samples for pharmacokinetic analysis will be taken on the first day of ALT-803 administration in the first study treatment cycle. Venous blood will be obtained at Time 0 (before the start of infusion), at 30 minutes, and 2, 4, 6 and 24 hours from Time 0 for the assessment of ALT-803 serum concentrations. Non-compartmental and compartmental analyses will be conducted. In addition, the same blood samples collected for PK analysis will be used to assess the serum levels of IL-2, IL-4, IL-6, IL-10, IFN- $\gamma$  and TNF- $\alpha$ . Fresh blood samples for immune cell levels and phenotype testing will be collected before the start of first and fourth dose of study drug infusion in each treatment cycle. Bone marrow samples will be collected for future analysis of molecular markers associated with responses or resistance to ALT-803 in patients with relapsed or refractory multiple myeloma.

#### **Monitoring Tests:**

Blood samples for standard chemistry and CBC with differential will be obtained at screening, on each study drug infusion day, and at follow-up visits. Blood samples for immunogenicity testing for anti-ALT-803 antibodies will be collected prior to dosing on the first ALT-803 infusion day, at week 7 and at the first assessment during week 11-12 from the initial dose of study treatment. Blood and urine samples will be collected on each follow-up visit for response assessment.

### Response Assessment:

There are at least two response assessments for treated patients: the first assessment during week 11-12 and the second assessment during week 23-24 from the start of study treatment. After completion of the first two cycles of study treatment, patients who have received at least 3 doses of study drug will have the first response assessment. After completion of the two additional cycles of study treatment, patients, regardless of the number of additional study drug doses received, will have the second response assessment. Response assessments will be carried out according to the new International Uniform Response Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. Baseline evaluations should be performed up to 14 days before study treatment starts.

### **Progression &**

#### Survival

**Assessment:** 

Progression-free survival, overall survival, and duration of response of all treated patients will be assessed every three months during year 1 and then every 6 months during years 2 and 3 from the start of study treatment, or through the point designated as the end of the study follow up.

**Adverse Events:** 

All patients will be monitored and evaluated for clinical toxicities during the treatment period and queried at each follow-up visit for Adverse Events (AEs). Patients may volunteer information concerning AEs. All adverse events will be graded by using the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0), and logged in the patient Case Report Form. The study centers should report all Serious Adverse Events (SAEs) and all events that trigger patient's study treatment discontinuation to the sponsor via phone, fax or email (or a combination) no more than 24 hours after learning of the event. The sponsor will use the information to manage and coordinate the dose escalation, cohort expansion and patient enrollment. The sponsor will then inform all of the participating clinical sites of the current dose level and the number of patients to be enrolled at that level, or of any patient enrollment suspension via phone, fax or email within 24 hours of learning of the event. The study centers should report all other adverse events to the sponsor following the guidelines defined in the study protocol. All study drug related AEs that are both serious and unexpected will be reported to the FDA in an expedited manner in accordance with 21 CFR §312.32.

Statistical Plan:

For each cohort, all AEs will be tabulated and examined and all safety, pharmacokinetic and tumor response data will be evaluated. For estimation of duration of response and progression free survival, the Kaplan-Meier method will be used. P-values of  $\leq 0.05$  (two-sided) will be considered to indicate statistical significance.

#### 8. STUDY CALENDAR, CLINICAL PROCEDURES & TESTS

### 8.1 Study calendar

| TESTS & PROCEDURES | SCREEN/<br>BASELINE <sup>1</sup> | Т | REAT | | T | REST | | REAT!<br>CYCL! | | | 1 <sup>ST</sup> RESPONSE<br>ASSESSMENT | TREATMENT CYCLES<br>#3 AND #4 | 2 <sup>ND</sup> RESPONSE<br>ASSESSMENT | FOLLOW-UPS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | | | | 1 | | 2 | | 2 - | | | 3 | 4-5 | 6 | 9 12 18 24 30 36 |
| Study Week | | 1 | 2 | 3 | 4 | 5-6 | 7 | 8 | 9 | 10 | 11-12 | 13-22 | 23-24 | |
| Study Day | | 1 | 8 | 15 | 22 | 23-42 | 43 | 50 | 57 | 64 | 71-84 | 85-148 | 155-168 | $\pm 1$ week |
| Tolerance Window | | | +/- 2 | days | | 23-42 | | +/- 2 a | lays | | Any day | | Any day | |
| Medical history | X | | | | | | | | | | | 1 | | |
| Serum pregnancy test <sup>2</sup> | X | | | | | | | | | | | Follow Institution's | | |
| Complete physical exam | X | X | | | | | X | | | | X | standard of care (SOC) | X | |
| Vital signs, Weight, Height <sup>3</sup> , Cardiac & Lung function monitoring | X | X | X | X | X | | X | X | X | X | X | policy. If performed, follow the | X | |
| Concurrent medication | X | X | X | X | X | | X | X | X | X | X | same schedule as in the | X | |
| Adverse event assessment <sup>4</sup> | X | X | X | X | X | | X | X | X | X | X | first two cycles of study | X | |
| CBC with Differential <sup>13</sup> | X | X | X | X | X | R | X | X | X | X | X | treatment. | X | |
| Blood Chemistry <sup>13</sup> | X | X | X | X | X | E | X | X | X | X | X | | X | |
| EKG | X | $X^5$ | | | | E | X | | | | | | | |
| PFT only when clinically indicated | X | | | | | S | | | | | | | | |
| Response evaluation <sup>6</sup> | | | | | | Т | | | | | X | | X | |
| Serum quantitative immunoglobulins | X | | | | | | | | | | X | | X | |
| SPEP | X | | | | | P | | | | | X | | X | |
| UPEP-random | X | | | | | | | | | | X | | X | |
| SIFE | X | | | | | E | | | | | X | | X | |
| UIFE -random | X | | | | | R | | | | | X | | X | |
| Serum FLC assay <sup>6.1</sup> | X | | | | | | | | | | X | | X | |
| Bone marrow plasma cell percentage <sup>6.2</sup> | X | | | | | I | | | | | X | | X | |
| Bone marrow immunohistochemistry or immunofluorescence <sup>6,3</sup> | | | | | | 0 | | | | | X | | X | |
| Soft tissue plasmacytomas assessment <sup>6.4</sup> | | | | | | D | | | | | X | | X | |
| Disease & survival follow-up/post-therapies <sup>7</sup> | | | | | | | | | | | | | | X X X X X X |
| Immune cell levels & phenotype <sup>8,11</sup> | | $X^8$ | | | $X^8$ | | $X^8$ | | | $X^8$ | | | | |
| PK <sup>12</sup> , IL-2, IL-4, IL-6, IL-10, IFN-γ, TNF- $\alpha^{9,11}$ | | $X^9$ | | | | | | | | | | | | |
| Immunogenicity tests <sup>10, 11</sup> | | $X^{10}$ | | | | | X | | | | X | | | |
| Study drug (ALT-803) | | a1 | a2 | а3 | a4 | | a5 | a6 | a7 | a8 | | Follow the same schedule as in the first 2 cycles of study treatment | | |

Screening/baseline evaluations are performed ≤ 14 days prior to start of therapy. If the patient's condition is deteriorating, ECOG status and laboratory evaluations should be repeated within 48 hours prior to initiation of study treatment infusion. <sup>2</sup>Pregnancy test is for women with childbearing potential only. <sup>3</sup>Vital signs (especially blood pressure), clinical status and laboratory tests should be reviewed before start of therapy. Day 1 for the 1<sup>st</sup> patient of each cohort will have vital signs evaluated at 15, 30, 60 and 120 min then hourly for 6 hours post infusion and every 3 hours thereafter until discharge (24 hrs). Vital signs for the rest of the study visits and all visits for subsequent patients will be evaluated at 15, 30, 60 and 120 min and then hourly post infusion until discharge (or at completion of dose monitoring) from the clinic. Body weight will be collected before infusion on each drug infusion day for all patients. <sup>4</sup>Patients who have an on-going study drug-related SAE upon study completion or at discontinuation of study will be contacted by the investigator or his/her designee every week until the event is resolved or determined to be irreversible. <sup>5</sup>If the screening EKG was performed within 14 days prior to start of study treatment, the EKG is not required. <sup>6</sup>Disease response and progression assessment will be evaluated using the new International Uniform Response Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. <sup>6,1</sup>Only when serum and urine M-protein and serum FLC are unmeasurable and bone marrow plasma cell percentage > 30% at baseline. <sup>6,3</sup>Only when scrim and urine M-protein and serum FLC are unmeasurable and bone marrow plasma cell percentage > 30% at baseline. <sup>6,4</sup>Only when scrim and urine M-protein and serum flow of tumor assessment & other therapies received after completion of study treatment will be collected if available. <sup>8</sup>Fresh blood samples for immune cell levels & phenotype testing will be collected before dosing. <sup>9</sup>Collect blood

<sup>&</sup>lt;sup>12</sup>The last PK sample will be collected on the next day. <sup>13</sup>Safety labs can be drawn within 24 hours of scheduled dose.

#### **CLINICAL STUDY PROTOCOL**

**Protocol Number:** CA-ALT-803-02-13

**Protocol Title:** A Study of ALT-803 in Patients with Relapsed

or Refractory Multiple Myeloma

**Date of Protocol:** 

 Version# 01
 January 7, 2014

 Version# 02
 February 3, 2014

 Version# 03
 February 5, 2014

 Version# 04
 May 16, 2014

 Version# 05
 December 17, 2015

Sponsor Contact: Alter BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

### **Table of Contents**

| S | YNOPS | IS | 6 |
|---|---|---|---|
| 1. | OBJ | ECTIVES | 12 |
| | 1.1 | PRIMARY OBJECTIVES | 12 |
| | 1.2 | SECONDARY OBJECTIVES | 12 |
| 2. | BAC | CKGROUND | 12 |
| | 2.1 | ALT-803 – General information | 12 |
| | 2.2 | MULTIPLE MYELOMA | |
| | 2.3 | IMMUNE-BASED THERAPIES FOR CANCER | |
| | 2.4 | PHARMACOLOGICAL EFFECTS OF ALT-803 IN VITRO AND IN ANIMALS | 14 |
| | 2.4.1 | | |
| | 2.4.2 | | |
| | 2.4.3<br>2.4.4 | 8 , 3 | |
| | 2.4.4 | | |
| | 2.5 | Non-clinical toxicology | |
| | 2.5.1 | | |
| | 2.5.2 | • | |
| | 2.6 | COMPARATIVE STUDIES OF INTRAVENOUS AND SUBCUTANEOUS ALT-803 | 19 |
| | 2.7 | PHARMACOKINETICS | |
| | 2.7.1 | 1 | |
| | 2.8 | RATIONALE FOR HUMAN CLINICAL STARTING DOSE | |
| | 2.9 | HUMAN EXPERIENCE | |
| 3. | RAT | TIONALE FOR THE CURRENT STUDY | 24 |
| 4. | OVI | ERALL STUDY DESIGN | 25 |
| 5. | STU | DY POPULATION | 26 |
| | 5.1 | INCLUSION CRITERIA | 26 |
| | 5.2 | EXCLUSION CRITERIA | 27 |
| | 5.3 | INCLUSION OF WOMEN AND MINORITIES | 27 |
| 6. | STU | DY DESIGN | 28 |
| | 6.1 | STUDY FLOW DIAGRAM | 28 |
| | 6.2 | SCREENING AND ENROLLMENT | 28 |
| | 6.3 | STUDY TREATMENT | |
| | 6.3.1 | - · | |
| | 6.3.2 | | |
| | 6.3.3<br>6.3.4 | Study drug preparation | |
| | 6.3.5 | | |
| | 6.4 | DURATION OF PATIENT PARTICIPATION | |
| | 6.5 | DOSE ESCALATION PHASE | |
| | 6.6 | EXPANSION PHASE | |
| | 6.7 | STOPPING RULES | |
| | 6.7.1 | During dose escalation phase of the study | 35 |
| | 6.7.2 | | |
| | 6.7.3 | | |
| | 6.8 | PATIENT MONITORING, RESPONSE EVALUATION, TREATMENT CYCLE #3 AND #4, DISEAS | |
| | & SURV<br>6.8.1 | /IVAL FOLLOW-UP | |
| | 0.0.1 | 1 444014 114014401416 | |

| | 6.8.2 | Response evaluation. | |
|---|---|---|---|
| | 6.8.3 | Treatment cycle #3 & #4 | |
| | 6.8.4 | Disease progression and survival follow-up | |
| ( | 6.9 I | OSE LIMITING TOXICITY | |
| | 6.9.1 | Definition of dose limiting toxicity | |
| | 6.9.2 | Definition of maximum tolerated dose (MTD) | |
| | 6.9.3 | Definition of minimal efficacious dose (MED) | |
| ( | 6.10 S | TUDY TREATMENT DISCONTINUATION | 37 |
| | 6.10.1 | Study treatment discontinuation events | |
| | 6.10.2 | Replacement of participants | |
| | 6.10.3 | Follow-ups after treatment discontinuation | |
| | | .3.1. Discontinuation due to SAEs or on-going study drug related AEs | |
| | | .3.2. Discontinuation due to any other reasons | |
| ( | | TUDY TREATMENT INTERRUPTION | |
| | 6.11.1 | Kidney dysfunction | |
| | 6.11.2 | Hematological dysfunction | |
| | 6.11.3 | Hypotension | |
| | 6.11.4 | Allergic reactions and cytokine release syndrome/acute infusion reaction | |
| ( | | GENERAL SUPPORTIVE CARE GUIDELINES AND DRUG INTERACTION | |
| | 6.12.1 | Hypotension and capillary leak syndrome | |
| | 6.12.2 | Pulmonary dysfunction | |
| | 6.12.3 | Impaired kidney and liver functions | |
| | 6.12.4 | Infection | |
| | 6.12.5 | Fever and chills | |
| | 6.12.6 | Gastritis | |
| | 6.12.7 | Diarrhea, nausea and vomiting | |
| | 6.12.8 | Pruritus and dermatitis | |
| | 6.12.9 | Acidosis | |
| | 6.12.10<br>6.12.11 | | |
| | 6.12.11 | | |
| _ | | | |
| 7. | STUD | Y DRUG: AVAILABILITY, ACCOUNTABILITY, PACKAGING & LABELING | 43 |
| , | 7.1 <i>A</i> | VAILABILITY | 43 |
| , | 7.2 A | ACCOUNTABILITY | 43 |
| , | 7.3 F | ACKAGING | 43 |
| , | | ABELING | |
| | | Y CALENDAR, CLINICAL PROCEDURES & TESTS | |
| 8. | | | |
| | | TUDY CALENDAR | |
| | | ROCEDURE AND TESTS | |
| | 8.2.1 | Assays for immune cell levels and phenotype | |
| | 8.2.2 | Medical history & prior therapy | |
| | 8.2.3 | Pregnancy test | |
| | 8.2.4 | Physical examination | |
| | 8.2.5 | Vital signs, body weight & height | |
| | 8.2.6 | Cardiac assessment | |
| | 8.2.7 | Pulmonary function monitoring | |
| | 8.2.8 | Clinical blood tests | |
| | 8.2.9 | Disease assessment tests and procedures | |
| | 8.2.10<br>8.2.11 | Adverse event assessment | |
| | 8.2.12 | Response assessment | |
| | 8.2.13 | Pharmacokinetic (PK) testing | |
| | 8.2.14 | Biomarker assays for IL-2, IL-4, IL-6, IL-10, IFN-γ, MCP-1 and TNF-α | |
| | 8.2.15 | Immunogenicity tests - detection of anti-ALT-803 antibodies | |
| | 0.4.10 | Invitation Continuity today well-cultivity of with IIII OUJ WILLOUNICS | |

| P. MEASUREMENT OF EFFECT | 50 |
|-----------------------------------------------------------------|-----|
| 9.1 Measurable disease | 50 |
| 9.2 EFFECT ASSESSMENT SCHEDULE | 50 |
| 9.3 METHODOLOGY OF RESPONSE EVALUATION | 50 |
| 9.4 RESPONSE EVALUATION CRITERIA | |
| 9.5 DISEASE PROGRESSION EVALUATION CRITERIA | 52 |
| 10. STATISTICAL ANALYSIS | 53 |
| 10.1 Study objectives | 53 |
| 10.2 Sample size | 53 |
| 10.3 Data collection | |
| 10.4 Data analysis | |
| 10.4.1 Analysis of safety | |
| 10.4.2 Analysis of response | |
| 10.4.3 Pharmacokinetics | |
| 11. REGULATORY AND REPORTING REQUIREMENTS | |
| 11.1 ADVERSE EVENTS RECORDING, REPORTING AND COMMUNICATION | |
| 11.2 ADVERSE EVENT TERMINOLOGY AND DEFINITIONS | |
| 11.3 ADVERSE EVENT REPORTING PROCEDURES | |
| 11.4 ADVERSE EVENT EXPEDITED REPORTING GUIDELINES | |
| 11.5 SUBMISSION OF SERIOUS ADVERSE EVENT REPORTING | |
| 11.6 DATA REPORTING FORMS | |
| 11.7 REPORT /DATA SUBMISSION ADDRESS & CONTACT | |
| 11.8 PATIENT RECORDS, QUALITY ASSURANCE, RECORDS RETENTION | |
| 11.10 SPECIAL REGULATORY CONSIDERATIONS | |
| 11.10 SPECIAL REGULATORY CONSIDERATIONS | |
| 11.10.2 Protocol amendments, informed consent, and IRB approval | 59 |
| 12. CONFIDENTIALITY | |
| 13. ETHICAL STANDARDS & INVESTIGATOR OBLIGATIONS | |
| 14. LIST OF EXPECTED ADVERSE EVENTS | |
| 15. CTCAE | |
| REFERENCES | |
| APPENDIX A: ECOG | |
| APPENDIX B: NEW YORK HEART ASSOCIATION CLASSIFICATION | |
| APPENDIX C: ETHICAL STANDARDS | |
| APPENDIX D: INVESTIGATOR OBLIGATIONS | |
| APPENDIX E: CONTACT LIST - ALTOR | |
| APPENDIX F: CONTACT LIST - DATA SAFETY MONITORING BOARD (DSMB) | |
| APPENDIX G: CONTACT LIST - LABORATORIES | |
| ALLENDIA U. CUNTACI LIST - LADUNATUNIES | / 4 |

#### **SYNOPSIS**

**Sponsor:** Altor Bioscience Corporation

**Protocol#:** CA-ALT-803-02-13

Study Drug Name: Not applicable

**Study Treatment** 

Active agents: ALT-803, a "recombinant human super agonist interleukin-15 (IL-15) complex"

(AKA, IL-15N72D:IL-15RαSu/IgG1 Fc complex)

**Study Type:** Interventional

**Study Phase:** I/II

**Protocol Title:** A Study of ALT-803 in Patients with Relapsed or Refractory Multiple Myeloma

**Objectives:** To evaluate the safety and tolerability of escalating doses, identify the Maximum

Tolerated Dose level (MTD) or Minimum Efficacious Dose (MED) and designate a dose level for Phase II study (RP2D) of ALT-803 in patients with relapsed or

refractory multiple myeloma.

To evaluate the effect of ALT-803 on the peripheral absolute lymphocyte counts (ALC) and white blood cell (WBC) counts, the number and phenotype of

peripheral blood T (total and subsets) and NK cells.

To estimate the anti-tumor activity of ALT-803 by radiologic or pathologic disease

response, progression free survival, and overall survival in treated patients.

To characterize the immunogenicity and pharmacokinetic profile, including serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ, MCP-1 and TNF-α, of ALT-803 in treated

patients.

**Study Design:** 

This is a Phase I/II, open-label, multi-center, competitive enrollment, and dose-escalation study of ALT-803 in patients with relapsed or refractory multiple myeloma.

The study includes a dose escalation phase to determine the MTD or MED using a modified classic (3+3) dose escalation design and to designate a dose level for the Phase II expansion phase (RP2D) and a two-stage expansion phase at the RP2D using a Simon two-stage design. In Phase I, seven cohorts will be evaluated. A step-down dose level (cohort# -1) will be provided in the event of encountering DLT in two patients at the planned initial dose level. In the absence of unacceptable toxicity or disease progression, each enrolled patient will receive up to four 6-week study treatment cycles, each consisting of a 4-week treatment period and a 2-week rest period. In each cycle for cohort 1, 2, 3 and 4, patients will receive four doses of ALT-803 by intravenous (IV) injection weekly for 4 weeks followed by a 2-week rest period. In each cycle for cohort 5, 6and 7 patients will receive four doses of ALT-803 by subcutaneous (SubQ) injection weekly for 4 weeks followed by a 2-week rest period. Patients with sufficient recovery of toxicities from the previous treatment cycles will be eligible to continue study treatment. After receiving two treatment cycles, patients who have at least stable

disease assessed at week 11-12 may receive up to two additional study treatment cycles followed by reassessment for continued tumor response.

The study will be conducted in conformity with Good Clinical Practice (GCP).

#### **Treatments:**

The study treatment plan for each enrolled patient includes up to four 6-week study treatment cycles. In each cycle for cohort 1, 2, 3 and 4 patients will receive four weekly doses of ALT-803 by intravenous injection followed by a 2-week rest period. In each cycle for cohort 5, 6 and 7 patients will receive four doses of ALT-803 by subcutaneous injection weekly for 4 weeks followed by a 2-week rest period. The rest period may be extended to include up to four additional weeks if necessary. Patients who do not experience or who sufficiently recover from toxicities of the previous treatment cycles will be eligible to continue the treatment included in the study treatment plan.

Treated patients will have up to two anti-tumor evaluation visits. Patients who receive at least three study drug doses during the first 2-cycle treatment period will be evaluated for anti-tumor response during week 11-12. Patients who have at least stable disease from the first anti-tumor evaluation and who meet other criteria to continue study treatment will receive up to two additional study treatment cycles, with the same treatment schedule, route of administration, and at the same dose level as the first two cycles; followed by reassessment for continued tumor response.

The study treatment and response evaluation visits are illustrated below (refer to study calendar for all study visits):

| Treatment Cycle Cycle | | | | | REST | | Cycl | le #2 | | Response<br>Evaluation | | Cycl | le #3 | | REST | Cycle #4 | | | | Response<br>Evaluation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Week | 1 | 2 | 3 | 4 | 5-6 | 7 | 8 | 9 | 10 | 11-12 | 13 | 14 | 15 | 16 | 17-18 | 19 | 20 | 21 | 22 | 23-24 |
| Treatment Day | 1 | 8 | 15 | 22 | 23-42 | 43 | 50 | 57 | 64 | 71-84 | 85 | 92 | 99 | 106 | 107-126 | 127 | 134 | 141 | 148 | 155-168 |
| Dose# | 1 | 2 | 3 | 4 | | 5 | 6 | 7 | 8 | | 9 | 10 | 11 | 12 | | 13 | 14 | 15 | 16 | |
| Response Evaluation | | | | | Rest<br>weeks | | | | | X | | | | | Rest<br>weeks | | | | | X |
| ALT-803 | X | X | X | X | | X | X | X | X | | X | X | X | X | | X | X | X | X | |

There are no restrictions on further therapies, such as chemotherapy, radiation therapy or surgery to be used after the protocol-specified therapy. Clearly, post-study treatments could be of significant clinical benefit in selected patients, and these patients will be followed for outcome.

Enrolled patients will receive the study treatment at qualified cancer treatment centers with adequate diagnostic and treatment facilities to provide appropriate management of therapy and complications. ALT-803 will be administered by intravenous infusion for cohort 1, 2, 3 and 4 into a central or peripheral vein under the supervision of a qualified physician experienced in the use of biologic anticancer agents. ALT-803 will be administered by subcutaneous injection for cohort 5, 6 and 7 under the supervision of a qualified physician experienced in the use of biologic anti-cancer agents.

# **Dose Escalation Phase:**

A modified 3 + 3 design will be used for identifying a tolerable dose for phase II studies by monitoring patients for DLTs to determine the MTD and for identifying an efficacious dose by monitoring patients' ALC and WBC count to determine the MED during the DLT observation period. The dose escalation phase is concluded when either the MTD or the MED is determined. A dose level (RP2D) will then be designated for Phase II study. There are seven cohorts of ALT-803 and a step-down cohort (-1) with a lower dose level of ALT-803 in the event that unexpected toxicity is encountered at the initial dose level.

Below are the planned dose levels and respective route of administration for the study drug during the dose escalation phase of the study.

| Cohort | ALT-803 Dose<br>(µg/kg) | Route | Number of patients |
|-------------|-------------------------|-------|--------------------|
| -1 | 0.5 | IV | 3 to 6 |
| 1 (initial) | 1 | IV | 3 to 6 |
| 2 | 3 | IV | 3 to 6 |
| 3 | 6 | IV | 3 to 6 |
| 4 | 10 | IV | 3 to 6 |
| 5 | 10 | SubQ | 3 to 6 |
| 6 | 15 | SubQ | 3 to 6 |
| 7 | 20 | SubQ | 3 to 6 |

Dose limiting toxicity (DLT) is defined as follows: any toxicity that is not clearly unrelated to drug administration that is of Grade 3 and does not resolve to Grade 1 or lower within a week despite the use of medical intervention or that is of Grade 4, with exceptions described in the study protocol.

The DLT Observation Period is defined as the duration of the first treatment cycle.

Maximum Tolerated Dose level (MTD) is defined as a dose level at which <2 out of 6 patients experienced DLT and that is one level below a dose that was not tolerated.

Minimal Efficacious Dose (MED) is defined as a dose level which produces an ALC  $\geq$ 25,000/µL sustained for 14 days or a total WBC  $\geq$ 35,000/µL sustained for 14 days among 2/3 or 4/6 of patients. For safety, we have also defined an "exceeding MED" as the occurrence of ALC  $\geq$ 35,000/µL or WBC  $\geq$ 50,000/µL sustained for 14 days.

# **Expansion Phase**

The two-stage expansion phase at the MTD or the MED level will be conducted using an optimal Simon's two-stage design. Objective response (OR) (defined as complete response (CR) + partial response (PR)) will be evaluated and set

thresholds of lack of efficacy (OR rate (ORR) = 10%) and an efficacy level of interest (ORR = 30%) will be selected.

### **Stopping Rules:**

Patient enrollment will be temporarily suspended based on occurrence of any of the following events, and the study committee, including the sponsor, the Data Safety Monitoring Board, and principal investigators will meet to discuss how to proceed with future patient enrollment in the study.

During the dose escalation phase of the study,

- If the maximum planned dose level has been reached, but neither the MTD nor MED can be determined.
- If de-escalation occurs and the step-down dose level cannot be designated as the MTD or MED.

Any time during the expansion phase of the study,

- More than 33% of patients experience a possible, probable or definite study drug related DLT.
- Favorable anti-tumor response data collected from enrolled patients.

At any time during the study,

The study committee may meet to discuss how to proceed with the study and may make any or all of the following recommendations for further patient enrollment:

- Downward adjustment of the study drug dose.
- Adjust the study drug dosing schedule.
- Recommend more effective pre-therapy, intra-therapy, and post-therapy side effect mitigation interventions.
- Correct protocol technical errors that caused unnecessary dose omissions or premature treatment discontinuations. After correction of protocol errors, the DSMB may meet to re-evaluate the safety profile of the study treatment and recommend how to proceed with the study, if necessary.

#### **Evaluations:**

Patients will be evaluated for clinical toxicities during the treatment. Patients' blood samples will be collected to assess the pharmacokinetic profile and immunogenicity of the study drug. The anti-tumor response will be evaluated at week 11-12 and week 23-24 from the start of study treatment. All patients who receive at least 3 doses of the study drug ALT-803 will be included in the anti-tumor response evaluation.

#### **Population:**

Patients of 18 years of age and above with relapsed or refractory multiple myeloma. Patients also need to have adequate cardiac, pulmonary, liver and kidney functions and have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

#### **Sample Size:**

A total of up to 42 assessable patients will be accrued to the dose escalation phase of the study (Phase I). Anticipated enrollment to this phase is 24 patients. Up to an additional 23 assessable patients will be enrolled at the expansion phase (Stage 1 and 2) of the study (Phase II). An estimated total of approximately 47 assessable patients will be enrolled to complete the study. Assuming a 20% rate of ineligible

or non-assessable cases, an estimated total of up to 57 patients may be accrued to the study.

# Primary Endpoints

#### For Phase I only

(1) Determination of the MTD or MED and designation of the recommended dose level (RP2D) for Phase II study of ALT-803 in patients with relapsed or refractory multiple myeloma.

#### For Phase I & II

- (2) Safety profile of ALT-803 in treated patients.
- (3) Disease response rate of treated patients.

# **Secondary Endpoints**

- (1) Evaluation of the effect of ALT-803 on the peripheral ALC and WBC counts, the number and phenotype of peripheral blood T (total and subsets) and NK cells in treated patients.
- (2) Duration of response in treated patients.
- (3) Progression free survival of treated patients.
- (4) Overall survival of treated patients.
- (5) Characterization of the immunogenicity and pharmacokinetic profile, including serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ, MCP-1 and TNF-α, of ALT-803 in treated patients.

### Pharmacokinetics & Biomarkers:

Fresh blood samples will be collected to assess immune cell levels and phenotype. Serum samples will be collected for pharmacokinetics and immunogenicity of the study drug ALT-803. The same serum samples collected for PK analysis will be used to assess the serum levels of IL-2, IL-4, IL-6, IL-10, IFN-γ, MCP-1, and TNF-α. Non-compartmental and compartmental PK analyses will be conducted. Bone marrow samples will be collected for future analysis of molecular markers associated with responses or resistance to ALT-803 in patients with relapsed or refractory multiple myeloma.

### **Monitoring Tests:**

Blood samples for standard chemistry and CBC with differential will be obtained at screening, on each study treatment day, and at follow-up visits. Blood samples for immunogenicity testing for anti-ALT-803 antibodies will be collected prior to dosing on the first ALT-803 treatment day, at week 7 and at the first assessment during week 11-12 from the initial dose of study treatment. Blood and urine samples will be collected on each follow-up visit for response assessment.

## Response Assessment:

There are at least two response assessments for treated patients: the first assessment during week 11-12 and the second assessment during week 23-24 from the start of study treatment. After completion of the first two cycles of study treatment, patients who have received at least 3 doses of study drug will have the first response assessment. After completion of the two additional cycles of study treatment, patients, regardless of the number of additional study drug doses received, will have the second response assessment. Response assessments will be carried out according to the new International Uniform Response Criteria for

Multiple Myeloma proposed by the International Myeloma Working Group. Baseline evaluations should be performed up to 28 days before study treatment starts.

# Progression & Survival Assessment:

Progression-free survival, overall survival, and duration of response of all treated patients will be assessed every three months during year 1 and then every 6 months during years 2 and 3 from the start of study treatment, or through the point designated as the end of the study follow up.

#### **Adverse Events:**

All patients will be monitored and evaluated for clinical toxicities during the treatment period and queried at each follow-up visit for Adverse Events (AEs). Patients may volunteer information concerning AEs. All adverse events will be graded by using the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0), and logged in the patient Case Report Form. The study centers should report all Serious Adverse Events (SAEs) and all events that trigger patient's study treatment discontinuation to the sponsor via phone, fax or email (or a combination) no more than 24 hours after learning of the event. The sponsor will use the information to manage and coordinate the dose escalation, cohort expansion, and patient enrollment. The sponsor will then inform all of the participating clinical sites of the current dose level and the number of patients to be enrolled at that level, or of any patient enrollment suspension via phone, fax, or email within 24 hours of learning of the event. The study centers should report all other adverse events to the sponsor following the guidelines defined in the study protocol. All study drug related AEs that are both serious and unexpected will be reported to the FDA in an expedited manner in accordance with 21 CFR §312.32.

#### **Statistical Plan:**

For each cohort, all AEs will be tabulated and examined and all safety, pharmacokinetic and tumor response data will be evaluated. For estimation of duration of response and progression free survival, the Kaplan-Meier method will be used. P-values of  $\leq 0.05$  (two-sided) will be considered to indicate statistical significance.

#### 8. STUDY CALENDAR, CLINICAL PROCEDURES & TESTS

### 8.1 Study calendar

| TESTS & PROCEDURES | SCREEN/<br>BASELINE <sup>1</sup> | | | TRI | EATM | IENT | CYC | LE #1 | l | | REST | | CYC | | | 1 <sup>ST</sup> RESPONSE<br>ASSESSMENT | TREATMENT<br>CYCLES<br>#3 AND #4 | 2 <sup>ND</sup> RESPONSE<br>ASSESSMENT | FOLLOW-UPS |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Month | | | | | | 1 | | | | | 2 | | 2 | - 3 | | 3 | 4-5 | 6 | 9 12 18 24 30 36 |
| Study Week | | | | • | | 2 | | | 4 | | 5-6 | 7 | 8 | 9 | 10 | 11-12 | 13-22 | 23-24 | |
| Study Day | | 1 | 2 | 3 | 4 | 8 | 15 | 22 | 23 | 25 | 23-42 | 43 | 50 | 57 | 64 | 71-84 | 85-148 | 155-168 | $\pm 1$ week |
| Tolerance Window | | | | | + | -/- 2 de | ays | | | | 23-42 | | +/- 2 | days days | | +/- 7 days | | +/- 7 days | |
| Medical history | X | | | | | | | | | | | | | | | | | | |
| Serum pregnancy test <sup>2</sup> | X | | | | | | | | | | | | | | | | Follow | | |
| Complete physical exam | X | X | | | | | | | | | | X | | | | X | Institution's | X | |
| Vital signs, Weight, Height <sup>3</sup> , Cardiac & Lung function monitoring | X | X | | | | X | X | X | | | | X | X | X | X | Х | standard of care<br>(SOC) policy. | X | |
| Concurrent medication | X | X | | | | X | X | X | | | | X | X | X | X | X | If performed, | X | |
| Adverse event assessment <sup>4</sup> | X | X | | | | X | X | X | | | | X | X | X | X | X | follow the same | X | |
| CBC with Differential <sup>12</sup> | X | X | | | | X | X | X | | | | X | X | X | X | X | schedule as in the | X | |
| Blood Chemistry <sup>12</sup> | X | X | | | | X | X | X | | | R | X | X | X | X | X | first two cycles of study treatment. | X | |
| EKG | X | $X^5$ | | | | | | | | | E | X | | | | | study treatment. | | |
| PFT only when clinically indicated | X | | | | | | | | | | s | | | | | | | | |
| Response evaluation <sup>6</sup> | | | | • | | | • | | | | | | • | • | - | X | | X | |
| Serum quantitative immunoglobulins | X | | | | | | | | | | T | | | | | X | | X | |
| SPEP | X | | | | | | | | | | | | | | | X | | X | |
| UPEP-random | X | | | | | | | | | | P | | | | | X | | X | |
| SIFE | X | | | | | | | | | | E | | | | | X | | X | |
| UIFE -random | X | | | | | | | | | | _ | | | | | X | | X | |
| Serum FLC assay <sup>6.1</sup> | X | | | | | | | | | | R | | | | | X | | X | |
| Bone marrow plasma cell percentage <sup>6.2</sup> | X | | | | | | | | | | I | | | | | X | | X | |
| Bone marrow immunohistochemistry or immunofluorescence <sup>6,3</sup> | | | | | | | | | | | 0 | | | | | Х | | X | |
| Soft tissue plasmacytomas assessment <sup>6,4</sup> | | | | | | | | | | | D | | | | | X | | X | |
| Disease & survival follow-up/post-therapies <sup>7</sup> | | | | | | | | | | | D | | | | | | | | X X X X X X |
| Immune cell levels & phenotype <sup>8,11</sup> | | $X^8$ | X | $X^{13}$ | X | | | $X^8$ | X | X | | $X^8$ | | | $X^8$ | | | | |
| PK, IL-2, IL-4, IL-6, IL-10, IFN- $\gamma$ , MCP-1 TNF- $\alpha^{9,11}$ | | X <sup>9</sup> | | $X^{13}$ | X | | | | | | | | | | | | | | |
| Immunogenicity tests <sup>10, 11</sup> | | $X^{10}$ | | | | | | | | | | X | | | | X | | | |
| Study drug (ALT-803) | | a1 | | | | a2 | a3 | a4 | | | | a5 | a6 | a7 | a8 | | Follow the same schedule as in the first 2 cycles | | |

Screening/baseline evaluations are performed  $\leq$  28 days prior to start of therapy. If the patient's condition is deteriorating, ECOG status and laboratory evaluations should be repeated within 48 hours prior to dosing.

Pregnancy test is for women with childbearing potential only. <sup>3</sup>Vital signs (especially blood pressure), clinical status and laboratory tests should be reviewed before start of therapy. Day 1 for the 1st patient of cohort 1, 2, 3 and 4 will have vital signs evaluated at 15, 30, 60 and 120 min then hourly for 6 hours post infusion and every 3 hours thereafter until discharge (24 hrs). Vital signs for subsequent patients and dosing visits in cohort 5, 6 and 7, vital signs will be evaluated at 15, 30, 60 and 120 min and then hourly post treatment until discharge (or at completion of dose monitoring) from the clinic. Body weight will be collected before treatment on each treatment day for all patients. <sup>4</sup>Patients who have an on-going study drug-related SAE upon study completion or at discontinuation of study will be contacted by the investigator or his/her designee every week until the event is resolved or determined to be irreversible. <sup>5</sup>If the screening EKG was performed within 28 days prior to start of study treatment, the EKG is not required. <sup>6</sup>Disease response and progression assessment will be evaluated using the new International Uniform Response Criteria for Multiple Myeloma proposed by the International Myeloma Working Group. <sup>6,1</sup>Only when serum and urine M-protein and serum FLC are unmeasurable and bone marrow plasma cell percentage > 30% at baseline. <sup>6,3</sup>Only when sex is to be determined. <sup>6,4</sup>Only when present at baseline, and to confirm CR or PR by X-rays, MRI or CT scans. <sup>7</sup>Information about tumor assessment & other therapies received after completion of study treatment will be collected if available. <sup>8</sup>Fresh blood samples for immune cell levels & phenotype testing will be collected before dosing. <sup>9</sup>Collect blood samples at Time 0 (before treatment), at 30 min (+/- 5 min), 2

IL-6, IL-10, IFN-γ, MCP-1 and TNF-α assays are performed using the same samples as PK. <sup>10</sup>Use the sample collected before dosing for PK test. <sup>11</sup>Residual samples may be used by Sponsor for research studies of other biomarkers. All attempts will be made to collect research samples but missed samples will not be considered a protocol deviation. <sup>12</sup>Safety labs can be drawn within 72 hours of scheduled dose. <sup>13</sup>The Cycle 1 Day 3 visit is optional if patient is available.